CLINICAL TRIAL: NCT03327571
Title: An International, Multi-centre, Non-interventional Retrospective Study to Describe Treatment Pathways, Outcomes, and Resource Use in Patients With Classical Hodgkin Lymphoma (B-HOLISTIC)
Brief Title: B-CD30 + Hodgkin Lymphoma International Multi-center Retrospective Study of Treatment Practices and Outcomes
Acronym: B-HOLISTIC
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: CHL-5001
Record Dates: First submitted 2017-10-27; First posted 2017-10-31 (Actual); Results first posted 2021-06-25 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: Classical Hodgkin Lymphoma; Relapsed or Refractory Classical Hodgkin Lymphoma
Keywords: Drug therapy
MeSH Terms: conditions — Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: cHL: Participants diagnosed with high-risk stage IIb-IV cHL, received frontline treatment with chemotherapy with or without radiotherapy between 01 January 2010 and 31 December 2013 from the 13 participating countries will be observed for various treatments received for cHL, associated adverse events and resources used from the date of cHL diagnosis until the date of first documented relapse or disease progression after frontline therapy. Participants will be continue to be observed for overall survival until the date of death or data collection, whichever occurs first.
- Group 2: RRHL: Participants diagnosed with RRHL, between 01 January 2010 and 31 December 2013 from the 13 participating countries will be observed for various treatments received for RRHL, detailed data on treatment pathways, clinical outcomes, associated adverse events and resources used from the date of RRHL diagnosis until the date death or data collection, whichever occurs first. Participants will be continue to be observed for overall survival until the date of death or data collection, whichever occurs first.

SUMMARY:
The purpose of this study is to describe progression-free survival (PFS) in participants with relapsed or refractory classical Hodgkin lymphoma (RRHL), defined as the time from initiation of first treatment for RRHL to first documentation of relapse or disease progression, or death.

DETAILED DESCRIPTION:
This is a retrospective, non-interventional study of participants with newly-diagnosed cHL, or with RRHL. The study will review the medical records of participants to describe participant's demographics, disease characteristics, treatments received, outcomes, health resources used by the participants, and adverse events that are associated with treatments, and resources used for treatment.

The study will enroll approximately 50 to 100 participants in each group at each of the 13 participating countries. Based on the diagnosis of the disease, participants will be assigned to one of the following groups:

Group 1: cHL Group 2: RRHL

This multi-center trial will be conducted in Argentina, Australia, China, Colombia, Hong Kong, Mexico, Republic of Korea, Russia, Saudi Arabia, Singapore, South Africa, Taiwan, and Turkey. The data for Group 1 and Group 2 will be collected from date of cHL or RRHL diagnosis until the date of death (or the date when the participant was last known to be alive, whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

1. Participants newly diagnosed with high-risk stage IIb-IV cHL (for Group 1) or RRHL (for Group 2) between 01 January 2010 and 31 December 2013.
2. Age greater than or equal to (>=) 18 years at diagnosis of cHL (Group 1) or RRHL (Group 2).
3. Alive or deceased.
4. Written informed consent is obtained for study data collection, where necessary, according to local regulations.

Exclusion Criteria:

1. Participants for whom the minimum study dataset is not available from their hospital medical records.
2. Participants who have participated in an interventional clinical trial at any stage of their cHL (Group 1) or RRHL (Group 2) management.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants diagnosed with high-risk stage IIb-IV cHL and/or with RRHL between 01 January 2010 and 31st December 2013 from the 13 participating countries.
Sampling Method: Non-Probability Sample
Enrollment: 1770 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Takeda
Locations (1):
- Pusan National University Hospital, Busan, South Korea

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Hernandez-Caballero A, Salazar R, Zerga M, Rivas-Vera S, Huang Z, Karduss A. Subgroup analysis of treatment pathways and clinical outcomes in Hodgkin lymphoma in Latin America from the retrospective B-HOLISTIC study. Sci Rep. 2025 Jul 7;15(1):24197. doi: 10.1038/s41598-025-07704-0. PMID 40624058
- [Derived] Ferhanoglu B, Kim TM, Karduss A, Brittain D, Tumyan G, Al-Mansour M, Zerga M, Song Y, Rivas-Vera S, Kwong YL, Lim ST, Yeh SP, Abdillah A, Huang Z, Dalal M, Wan H, Hertzberg M. Treatment pathways and clinical outcomes in Hodgkin lymphoma outside Europe and North America: results from the international, multicenter, retrospective, B-HOLISTIC study. Leuk Lymphoma. 2022 Dec;63(14):3317-3330. doi: 10.1080/10428194.2022.2126281. Epub 2022 Oct 6. PMID 36200380

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data abstraction took place in Argentina, Australia, China, Colombia, Hong Kong, Mexico, Russia, Saudi Arabia, South Africa, Province Of China, Turkey, Singapore and Republic of Korea from 21 November 2017 to 31 October 2019. Participants diagnosed with high-risk stage IIb-IV classical Hodgkin lymphoma (cHL) (Group 1) or with relapsed/refractory classical Hodgkin lymphoma (RRHL) (Group 2) between 2010 and 2013 were observed in this study.
Pre-assignment Details: 1770 participants were enrolled in this study, of which, 1703 were eligible for analysis set of the study. Out of 1703 participants, 1598 participants were eligible and enrolled in Group 1 (cHL) and further, 426 participants were eligible and enrolled in Group 2 (RRHL). Out of 426 participants in Group 2, 321 participants who were diagnosed with CHL, and subsequently RRHL between 2010 and 2013 were common in Group 1 and 2.
Groups:
- Group 1: cHL: Participants diagnosed with high-risk stage IIb-IV cHL between 01 January 2010 and 31 December 2013, who received frontline treatment with chemotherapy with or without radiotherapy, and participants who were diagnosed with high-risk stage IIb-IV cHL and then were subsequently diagnosed with RRHL between 2010 and 2013 were observed retrospectively until the date of death or data collection, whichever occurred first.
- Group 2: RRHL: Participants diagnosed with RRHL between 01 January 2010 and 31 December 2013, and participants who were diagnosed with high-risk stage IIb-IV cHL and then were subsequently diagnosed with RRHL between 2010 and 2013 were observed retrospectively until the date of death or data collection, whichever occurred first.
Period: Group 1: cHL
Arm/Group | Group 1: cHL | Group 2: RRHL
Started | 1598 | 0
Completed | 1598 | 0
Not Completed | 0 | 0
Period: Group 2: RRHL
Arm/Group | Group 1: cHL | Group 2: RRHL
Started | 0 | 426 (105 RRHL only participants and 321 common participants who had CHL, and subsequently RRHL between 2010-2013.)
Participants Were Counted in Both Groups | 0 | 321 (Participants who were diagnosed with CHL, and subsequently RRHL between 2010 and 2013.)
Completed | 0 | 426
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all participants who were eligible for cHL or RRHL group including the common participants in both the groups.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1: cHL | Group 2: RRHL | Total
Number analyzed (Participants) | 1598 | 105 | 1703
Age, Customized [Count of Participants; unit: Participants]
  Less than (<) 60 years | 1382 | 94 | 1476
  Greater than or equal to (>=) 60 years | 216 | 11 | 227
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 719 | 41 | 760
  Male | 879 | 64 | 943
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 62 | 2 | 64
  American Indian or Alaska Native | 22 | 0 | 22
  Asian | 560 | 29 | 589
  White or Caucasian | 525 | 57 | 582
  Not Reported | 197 | 12 | 209
  Other | 232 | 5 | 237

OUTCOME MEASURES:

1. Primary Outcome: Group 2, RRHL: Progression Free Survival (PFS)
Description: PFS was defined as time from initiation of frontline regimen to first documentation of relapse or disease progression or death, censored at date of most recent follow-up/contact. Progressive disease (PD) was defined as any new lesion or increase by >=50% of previously involved site from nadir, and was evaluated based on International Working Group (IWG) criteria (Cheson et al 2007). Median PFS was estimated using the Kaplan-Meier method.
Time Frame: From initiation of first treatment until first documentation of relapse/PD/until date of death (or date when participant was last alive), whichever occurred first (observed retrospectively from 2010 until date of data collection [up to 9 years 10 months])
Population: The FAS included all participants who were eligible for RRHL group including the common participants in both the groups.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 426
months | 13.17 [9.92 to 20.17]

2. Secondary Outcome: Group 1, cHL: Number of Participants Based on Clinical Staging According to Ann Arbor Staging at Diagnosis
Description: The Ann Arbor staging system of lymphomas is used to summarize the extent of the cancer's spread. Stages are classified by Roman numerals I (lessspread) to IV (more spread). Additional sub staging variables include: A, asymptomatic; and B, presence of B symptoms (including fever, night sweats and weight loss of >=10 percent [%] of body weight over 6 months).
Time Frame: Day 1 at cHL diagnosis
Population: The FAS included all participants who were eligible for cHL group including the common participants in both the groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: cHL
Number analyzed (Participants) | 1598
Participants
  Stage I-A | 0
  Stage I-B | 0
  Stage II-A | 0
  Stage II-B | 441
  Stage III-A | 207
  Stage III-B | 356
  Stage IV-A | 161
  Stage IV-B | 433
  Stage unknown | 0

3. Secondary Outcome: Group 2, RRHL: Number of Participants Based on Clinical Staging According to Ann Arbor Staging at Diagnosis
Description: The Ann Arbor staging system of lymphomas is used to summarize the extent of the cancer's spread. Stages are classified by Roman numerals I (lessspread) to IV (more spread). Additional sub staging variables include: A, asymptomatic; and B, presence of B symptoms (including fever, night sweats and weight loss of >=10 % of body weight over 6 months).
Time Frame: Day 1 at RRHL diagnosis
Population: The FAS included all participants who were eligible for RRHL group including the common participants in both the groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 426
Participants
  Stage I-A | 7
  Stage I-B | 2
  Stage II-A | 24
  Stage II-B | 61
  Stage III-A | 52
  Stage III-B | 78
  Stage IV-A | 53
  Stage IV-B | 107
  Stage unknown | 42

4. Secondary Outcome: Group 2, RRHL: Number of Participants Based on Clinical Staging According to Ann Arbor Staging at Relapse After First Relapse or Refractory Diagnosis
Description: The Ann Arbor staging system of lymphomas is used to summarize the extent of the cancer's spread. Stages are classified by Roman numerals I (less spread) to IV (more spread). Additional sub staging variables include: A, asymptomatic; and B, presence of B symptoms (including fever, night sweats and weight loss of >=10% of body weight over 6 months).
Time Frame: At second, third, fourth, and fifth relapse (up to 9 years 10 months)
Population: The FAS included all participants who were eligible for RRHL group including the common participants in both the groups. Here "overall number of participants" analyzed are those who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 79
Participants
  Clinical stage at 2nd relapse: Stage I-A | 1
  Clinical stage at 2nd relapse: Stage I-B | 0
  Clinical stage at 2nd relapse: Stage II-A | 6
  Clinical stage at 2nd relapse: Stage II-B | 9
  Clinical stage at 2nd relapse: Stage III-A | 9
  Clinical stage at 2nd relapse: Stage III-B | 15
  Clinical stage at 2nd relapse: Stage IV-A | 9
  Clinical stage at 2nd relapse: Stage IV-B | 14
  Clinical stage at 2nd relapse: Stage unknown | 16
  Clinical stage at 3rd relapse: number analyzed (Participants) | 22
  Clinical stage at 3rd relapse: Stage I-A | 0
  Clinical stage at 3rd relapse: Stage I-B | 0
  Clinical stage at 3rd relapse: Stage II-A | 2
  Clinical stage at 3rd relapse: Stage II-B | 4
  Clinical stage at 3rd relapse: Stage III-A | 2
  Clinical stage at 3rd relapse: Stage III-B | 4
  Clinical stage at 3rd relapse: Stage IV-A | 1
  Clinical stage at 3rd relapse: Stage IV-B | 3
  Clinical stage at 3rd relapse: Stage unknown | 6
  Clinical stage at 4th relapse: number analyzed (Participants) | 8
  Clinical stage at 4th relapse: Stage I-A | 1
  Clinical stage at 4th relapse: Stage I-B | 0
  Clinical stage at 4th relapse: Stage II-A | 1
  Clinical stage at 4th relapse: Stage II-B | 0
  Clinical stage at 4th relapse: Stage III-A | 0
  Clinical stage at 4th relapse: Stage III-B | 1
  Clinical stage at 4th relapse: Stage IV-A | 1
  Clinical stage at 4th relapse: Stage IV-B | 2
  Clinical stage at 4th relapse: Stage unknown | 2
  Clinical stage at 5th relapse: number analyzed (Participants) | 2
  Clinical stage at 5th relapse: Stage I-A | 0
  Clinical stage at 5th relapse: Stage I-B | 0
  Clinical stage at 5th relapse: Stage II-A | 1
  Clinical stage at 5th relapse: Stage II-B | 0
  Clinical stage at 5th relapse: Stage III-A | 0
  Clinical stage at 5th relapse: Stage III-B | 0
  Clinical stage at 5th relapse: Stage IV-A | 0
  Clinical stage at 5th relapse: Stage IV-B | 0
  Clinical stage at 5th relapse: Stage unknown | 1

5. Secondary Outcome: Group 1, cHL: Number of Participants Based on Each International Prognostic Score (IPS) Category
Description: IPS score was calculated based on following factors: age >=45 years, male sex, stage IV disease, albumin<4 gram per liter (g/L), white blood cell (WBC)>=15*10^9 per liter (/L), haemoglobin <10.5 g/L, and lymphocyte count<0.6*10^6/L or <8% of differential. One point was assigned for each of above factors. The sum of points allotted correlates with following risk groups: good risk (0-1 points)-5 year survival of 89-90%; fair risk (2 to 3 points)-5 year survival of 78-81%; poor risk (4-7 points)-5 year survival of 56-61%. Total score range is 0 to 7, lower scores indicate higher survival rate.
Time Frame: Day 1 at cHL diagnosis
Population: The FAS included all participants who were eligible for cHL group including the common participants in both the groups. Here "overall number of participants" analyzed are those who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: cHL
Number analyzed (Participants) | 1087
Participants
  Good risk (IPS 0-1) | 289
  Fair risk (IPS 2-3) | 504
  Poor risk (IPS 4-7) | 294

6. Secondary Outcome: Group 1, cHL: Number of Participants With B Symptoms at Diagnosis
Description: The Ann Arbor staging system of lymphomas is used to summarize the extent of the cancer's spread. Stages are classified by Roman numerals I (less spread) to IV (more spread). If the following symptoms (B-symptoms) are present, a "B" classification is added to the stage: fever, night sweats and weight loss of >=10% of body weight over 6 months. B-symptoms indicate the presence of systemic symptoms. The presence or absence of B-symptoms has prognostic significance and is reflected in the staging of these lymphomas.
Time Frame: Day 1 at cHL diagnosis
Population: The FAS included all participants who were eligible for cHL group including the common participants in both the groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: cHL
Number analyzed (Participants) | 1598
Participants
  Presence of B-symptoms | 1230
  Absence of B-symptoms | 368

7. Secondary Outcome: Group 2, RRHL: Number of Participants With B Symptoms at Diagnosis
Description: as for outcome 6
Time Frame: Day 1 at RRHL diagnosis
Population: The FAS included all participants who were eligible for RRHL group including the common participants in both the groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 426
Participants
  Presence of B-symptoms | 248
  Absence of B-symptoms | 178

8. Secondary Outcome: Group 2, RRHL: Number of Participants Categorized Based on Prior Therapies for Hodgkin Lymphoma (HL) at Each Line of Treatment
Description: Number of participants were categorized based on prior therapies for HL at each line of treatment.
Time Frame: Day 1 at RRHL diagnosis
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 425
Participants
  Frontline treatment | 425
  Second line treatment | 17
  Third line treatment | 1
  Pre-SCT line treatment | 1

9. Secondary Outcome: Group 2, RRHL: Median Number of Previous Treatment Regimens (Chemotherapies) Received
Time Frame: Day 1 at RRHL diagnosis
Population: as for outcome 4
Measure: Median (Full Range); unit: previous treatment regimen
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 425
previous treatment regimen | 1.0 [1.0 to 4.0]

10. Secondary Outcome: Group 1, cHL: Number of Participants Categorized Based on Frontline Treatment Regimens
Description: Therapy regimens were numbered as 1: Doxorubicin (Doxo) + Bleomycin (bleo) + Vinblastine (Vinbl) + Decarbazine (Dacar) (ABVD); 3: Doxo + Vinbl + Mechlorethamine + Etoposide (Eto) + Vincristilne (Vinc) + Bleo + Prednisone (Pred) (Stanford V); 6: Cyclophophamide (Cyclo) + Vinc + Procarbazine (Procarb) + Pred (C-MOPP); 7: Dexamethasone + Cytarabine + Cisplatin (DHAP); 8: Eto + Methylprednisolone + Cytarabine + Cisplatin (ESHAP); 10: Ifosfamide+ Carboplatin + Eto (ICE); 11: Ifosfamide + Gemcitabine +Vinorelbine + Pred (IGEV); 17: Rituximab; 18: Brentuximab vedotin; 4: Bleo + Eto + Doxo + Cyclo + Vinc + Procarb + Pred (BEACOPP); 14: Cycl + Doxo + Vinc + Pred (CHOP); 15: Cycl + Vinc + Pred (CVP); 2: ABVD + Doxo + Bleo + Vinbl + Dacar then Bleo + Eto + Doxo + Cycl + Vinc + Procarb+ Pred ( Escalated BEACOPP); 24: Other.
Time Frame: From initial diagnosis until the date of death (or the date when the participant was last known to be alive) (observed retrospectively from 2010 until date of data collection [up to 9 years 10 months])
Population: The FAS included all participants who were eligible for cHL group including the common participants in both the groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: cHL
Number analyzed (Participants) | 1598
Participants
  Therapy regimen 1 | 1363
  Therapy regimen 3 | 1
  Therapy regimen 6 | 2
  Therapy regimen 7 | 9
  Therapy regimen 8 | 11
  Therapy regimen 10 | 3
  Therapy regimen 11 | 1
  Therapy regimen 17 | 2
  Therapy regimen 18 | 1
  Therapy regimen 4 | 104
  Therapy regimen 14 | 15
  Therapy regimen 15 | 4
  Therapy regimen 2 | 33
  Therapy regimen 24 | 114

11. Secondary Outcome: Group 1, cHL: Median Number of Treatment Cycles Associated With Each Frontline Treatment Regimen
Description: Therapy regimens were numbered as 1: ABVD; 3: Stanford V; 6: C-MOPP; 7: DHAP; 8: ESHAP; 10: ICE; 11: IGEV; 17: Rituximab; 18: Brentuximab vedotin; 4: BEACOPP; 14: CHOP; 15: CVP; 2: ABVD + Escalated BEACOPP; 24: Other.
Time Frame: as for outcome 10
Population: The FAS included all participants who were eligible for cHL group including the common participants in both the groups. Here "overall number of participants" analyzed are those who were evaluable for this outcome measure. Here number analyzed "n" are the participants who were evaluable for the outcome measure at given categories.
Measure: Median (Full Range); unit: cycles
Arm/Group | Group 1: cHL
Number analyzed (Participants) | 1362
cycles
  Therapy regimen 1 | 6.0 [6.0 to 6.0]
  Therapy regimen 3: number analyzed (Participants) | 1
  Therapy regimen 3 | 5.0 [5.0 to 5.0]
  Therapy regimen 6: number analyzed (Participants) | 2
  Therapy regimen 6 | 6.0 [6.0 to 6.0]
  Therapy regimen 7: number analyzed (Participants) | 9
  Therapy regimen 7 | 2.0 [1.0 to 4.0]
  Therapy regimen 8: number analyzed (Participants) | 11
  Therapy regimen 8 | 2.0 [2.0 to 6.0]
  Therapy regimen 10: number analyzed (Participants) | 3
  Therapy regimen 10 | 2.0 [2.0 to 2.0]
  Therapy regimen 11: number analyzed (Participants) | 1
  Therapy regimen 11 | 4.0 [4.0 to 4.0]
  Therapy regimen 17: number analyzed (Participants) | 2
  Therapy regimen 17 | 7.0 [6.0 to 8.0]
  Therapy regimen 18: number analyzed (Participants) | 1.0
  Therapy regimen 18 | 3.0 [3.0 to 3.0]
  Therapy regimen 4: number analyzed (Participants) | 104
  Therapy regimen 4 | 6.0 [1.0 to 8.0]
  Therapy regimen 14: number analyzed (Participants) | 15
  Therapy regimen 14 | 6.0 [1.0 to 8.0]
  Therapy regimen 15: number analyzed (Participants) | 4
  Therapy regimen 15 | 3.5 [1.0 to 7.0]
  Therapy regimen 2: number analyzed (Participants) | 33
  Therapy regimen 2 | 6.0 [4.0 to 11.0]
  Therapy regimen 24: number analyzed (Participants) | 114
  Therapy regimen 24 | 6.0 [1.0 to 9.0]

12. Secondary Outcome: Group 1, cHL: Number of Participants Who Received Treatments for HL After Completion of Frontline Therapy (Before Relapse)
Description: Therapy regimens were numbered as 1: ABVD; 6: C-MOPP; 7: DHAP; 8: ESHAP; 10: ICE; 11: IGEV; 12: Carmustine + Cytarabine + Etoposide + Melphalan (Mini-BEAM); 13: Etoposide + Ifosfamide + Mesna + Mitoxantrone (MINE); 18: Brentuximab vedotin; 16: Gemcitabine + Vinoreilbine + Pegylated liposomal doxorubicin (GVD); 4: BEACOPP; 14: CHOP; 24: Other.
Time Frame: as for outcome 10
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: cHL
Number analyzed (Participants) | 63
Participants
  Therapy regimen 1 | 2
  Therapy regimen 6 | 1
  Therapy regimen 7 | 8
  Therapy regimen 8 | 15
  Therapy regimen 10 | 8
  Therapy regimen 11 | 6
  Therapy regimen 12 | 2
  Therapy regimen 13 | 1
  Therapy regimen 18 | 2
  Therapy regimen 16 | 6
  Therapy regimen 4 | 6
  Therapy regimen 14 | 2
  Therapy regimen 24 | 10

13. Secondary Outcome: Group 1, cHL: Number of Participants Based on Radiotherapy (RT) Type and Site When Received at Frontline
Time Frame: as for outcome 10
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: cHL
Number analyzed (Participants) | 409
Participants
  RT Type: Whole body | 10
  RT Type: Involved-field | 244
  RT Type: Involved-site | 94
  RT Type: Involved-node | 60
  RT Type: Other | 1
  RT Site: Abdominal nodes | 8
  RT Site: Axillary nodes | 21
  RT Site: Bone lesions | 9
  RT Site: Breast | 3
  RT Site: Cervix | 3
  RT Site: Inguinal nodes | 7
  RT Site: Larynx | 1
  RT Site: Lung | 5
  RT Site: Mediastinal nodes | 197
  RT Site: Neck nodes | 69
  RT Site: Pancreas | 1
  RT Site: Para-aortic nodes | 6
  RT Site: Para-iliac nodes | 3
  RT Site: Pelvic nodes | 7
  RT Site: Skin | 3
  RT Site: Soft tissue | 2
  RT Site: Spleen | 7
  RT Site: Supraclavicular nodes | 14
  RT Site: Thyroid | 1
  RT Site: Other | 42

14. Secondary Outcome: Group 1, cHL: Number of Participants Categorized Based on RT Treatment Given as Pre-planned Frontline Treatment and RT Treatment Given for Residual Fluorodeoxyglucose (FDG)-Avid Disease
Description: Assessment was done for RT's whether used for pre-planned frontline treatment or for residual Fluorodeoxyglucose (FDG)-avid disease.
Time Frame: as for outcome 10
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: cHL
Number analyzed (Participants) | 409
Participants
  RT for pre-planned frontline treatment | 225
  RT for residual FDG-avid disease | 115

15. Secondary Outcome: Group 2, RRHL: Percentage of Participants Categorized Based on ASCT Eligibility Assessment
Time Frame: as for outcome 10
Population: The FAS included all participants who were eligible for RRHL group including the common participants in both the groups. Here "overall number of participants" analyzed are those who were evaluable for this outcome measure. Here number analyzed "n" are the participants who were evaluable for the outcome measure at given categories.
Measure: Number; unit: percentage of participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 425
percentage of participants
  Eligible for ASCT | 68.7
  Ineligible for ASCT | 31.3
  Initially ineligible and became eligible for ASCT: number analyzed (Participants) | 131
  Initially ineligible and became eligible for ASCT | 7.6
  Became eligible and received ASCT: number analyzed (Participants) | 10
  Became eligible and received ASCT | 60.0
  Eligible and received ASCT: number analyzed (Participants) | 302
  Eligible and received ASCT | 73.5
  Eligible and did not receive ASCT: number analyzed (Participants) | 302
  Eligible and did not receive ASCT | 26.5

16. Secondary Outcome: Group 2, RRHL: Median Number of Treatment Cycles Associated With Relapse/ Refractory Treatment Regimen for ASCT
Description: Therapy regimens were numbered as 1: ABVD; 6: C-MOPP; 8: ESHAP; 11: IGEV; 12: Mini-BEAM; 18: Brentuximab vedotin; 22: Nivolumab; 24: Other.
Time Frame: as for outcome 10
Population: The FAS included all participants who were eligible for RRHL group including the common participants in both the groups. . Here "overall number of participants" analyzed are those who were evaluable for this outcome measure. Here number analyzed "n" are the participants who were evaluable for the outcome measure at given categories.
Measure: Median (Full Range); unit: cycles
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 6
cycles
  Therapy regimen 1 | 6.0 [1.0 to 8.0]
  Therapy regimen 6: number analyzed (Participants) | 1
  Therapy regimen 6 | 8.0 [8.0 to 8.0]
  Therapy regimen 8: number analyzed (Participants) | 3
  Therapy regimen 8 | 2.0 [2.0 to 4.0]
  Therapy regimen 11: number analyzed (Participants) | 3
  Therapy regimen 11 | 3.0 [2.0 to 3.0]
  Therapy regimen 12: number analyzed (Participants) | 1
  Therapy regimen 12 | 5.0 [5.0 to 5.0]
  Therapy regimen 18: number analyzed (Participants) | 2
  Therapy regimen 18 | 4.0 [4.0 to 4.0]
  Therapy regimen 22: number analyzed (Participants) | 1
  Therapy regimen 22 | 6.0 [6.0 to 6.0]
  Therapy regimen 24: number analyzed (Participants) | 5
  Therapy regimen 24 | 2.0 [2.0 to 16.0]

17. Secondary Outcome: Group 2, RRHL: Number of Non-ASCT Participants Categorized Based on Reasons for Not Undergoing ASCT Despite Being ASCT Eligible
Description: Reasons for ASCT-eligible participants for not undergoing ASCT included participant refusal, inability to mobilize stem cells, loss of response to chemotherapy, cumulative toxicities, comorbid conditions, others, and unknown.
Time Frame: as for outcome 10
Population: The FAS included all participants who were eligible for RRHL group including common participants. Here "overall number of participants" analyzed are those who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 80
Participants
  Participant refusal | 21
  Inability to mobilize stem cells | 3
  Loss of response to chemotherapy | 13
  Cumulative Toxicities | 1
  Other | 11
  Comorbid conditions | 2
  Unknown | 29

18. Secondary Outcome: Group 2, RRHL: Number of Non-ASCT Participants Based on Reasons for ASCT Ineligibility
Description: Reasons for ASCT ineligibility included advanced age, comorbid conditions, chemoresistant disease, cumulative toxicities, and others.
Time Frame: as for outcome 10
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 201
Participants
  Advanced age: number analyzed (Participants) | 121
  Advanced age | 12
  Comorbid conditions: number analyzed (Participants) | 121
  Comorbid conditions | 13
  Chemo-resistant disease: number analyzed (Participants) | 121
  Chemo-resistant disease | 19
  Cumulative toxicities: number analyzed (Participants) | 121
  Cumulative toxicities | 1
  Other: number analyzed (Participants) | 121
  Other | 11
  Participant refusal | 5
  Inability to mobilize stem cells | 1
  Loss of response to chemotherapy: number analyzed (Participants) | 121
  Loss of response to chemotherapy | 4
  Unknown: number analyzed (Participants) | 121
  Unknown | 55

19. Secondary Outcome: Group 2, RRHL: Number of Non-ASCT Participants Categorized Based on Treatment Regimens Received at Each Line of Treatment
Description: Therapy regimens were numbered as 1: ABVD; 2: ABVD followed by Escalated BEACOPP; 3: Stanford V; 4: BEACOPP; 6: Cyclophosphamide C-MOPP; 7: DHAP; 8: ESHAP; 9: GCD; 10: ICE; 11: IGEV; 12: Mini-BEAM; 13: MINE; 14: CHOP; 15: CVP; 16: GVD; 17: Rituximab; 18: Brentuximab vedotin; 19: Bendamustine; 22: Nivolumab; 23: Pembrolizumab; 24: Other. More than one line of treatment or therapy was selected for each participant.
Time Frame: as for outcome 10
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 201
Participants
  Frontline: Therapy regimen 1 | 161
  Frontline: Therapy regimen 3 | 1
  Frontline: Therapy regimen 6 | 1
  Frontline: Therapy regimen 7 | 4
  Frontline: Therapy regimen 11 | 1
  Frontline: Therapy regimen 18 | 1
  Front line: Therapy regimen 4 | 16
  Frontline: Therapy regimen 14 | 3
  Frontline: Therapy regimen 15 | 1
  Frontline: Therapy regimen 2 | 6
  Frontline: Therapy regimen 24 | 16
  Second line: Therapy regimen 1: number analyzed (Participants) | 157
  Second line: Therapy regimen 1 | 13
  Second line: Therapy regimen 6: number analyzed (Participants) | 157
  Second line: Therapy regimen 6 | 3
  Second line: Therapy regimen 7: number analyzed (Participants) | 157
  Second line: Therapy regimen 7 | 23
  Second line: Therapy regimen 8: number analyzed (Participants) | 157
  Second line: Therapy regimen 8 | 21
  Second line: Therapy regimen 9: number analyzed (Participants) | 157
  Second line: Therapy regimen 9 | 1
  Second line: Therapy regimen 10: number analyzed (Participants) | 157
  Second line: Therapy regimen 10 | 18
  Second line: Therapy regimen 11: number analyzed (Participants) | 157
  Second line: Therapy regimen 11 | 7
  Second line: Therapy regimen 13: number analyzed (Participants) | 157
  Second line: Therapy regimen 13 | 7
  Second line: Therapy regimen 17: number analyzed (Participants) | 157
  Second line: Therapy regimen 17 | 2
  Second line: Therapy regimen 18: number analyzed (Participants) | 157
  Second line: Therapy regimen 18 | 1
  Second line: Therapy regimen 19: number analyzed (Participants) | 157
  Second line: Therapy regimen 19 | 1
  Second line: Therapy regimen 4: number analyzed (Participants) | 157
  Second line: Therapy regimen 4 | 13
  Second line: Therapy regimen 14: number analyzed (Participants) | 157
  Second line: Therapy regimen 14 | 5
  Second line: Therapy regimen 15: number analyzed (Participants) | 157
  Second line: Therapy regimen 15 | 1
  Second line: Therapy regimen 2: number analyzed (Participants) | 157
  Second line: Therapy regimen 2 | 5
  Second line: Therapy regimen 24: number analyzed (Participants) | 157
  Second line: Therapy regimen 24 | 39
  Third line: Therapy regimen 1: number analyzed (Participants) | 64
  Third line: Therapy regimen 1 | 3
  Third line: Therapy regimen 7: number analyzed (Participants) | 64
  Third line: Therapy regimen 7 | 4
  Third line: Therapy regimen 8: number analyzed (Participants) | 64
  Third line: Therapy regimen 8 | 3
  Third line: Therapy regimen 9: number analyzed (Participants) | 64
  Third line: Therapy regimen 9 | 2
  Third line: Therapy regimen 10: number analyzed (Participants) | 64
  Third line: Therapy regimen 10 | 8
  Third line: Therapy regimen 11: number analyzed (Participants) | 64
  Third line: Therapy regimen 11 | 11
  Third line: Therapy regimen 13: number analyzed (Participants) | 64
  Third line: Therapy regimen 13 | 3
  Third line: Therapy regimen 17: number analyzed (Participants) | 64
  Third line: Therapy regimen 17 | 1
  Third line: Therapy regimen 18: number analyzed (Participants) | 64
  Third line: Therapy regimen 18 | 3
  Third line: Therapy regimen 22: number analyzed (Participants) | 64
  Third line: Therapy regimen 22 | 1
  Third line: Therapy regimen 4: number analyzed (Participants) | 64
  Third line: Therapy regimen 4 | 2
  Third line: Therapy regimen 24: number analyzed (Participants) | 64
  Third line: Therapy regimen 24 | 23
  Other treatment: Therapy regimen 6: number analyzed (Participants) | 24
  Other treatment: Therapy regimen 6 | 1
  Other treatment: Therapy regimen 7: number analyzed (Participants) | 23
  Other treatment: Therapy regimen 7 | 1
  Other treatment: Therapy regimen 10: number analyzed (Participants) | 23
  Other treatment: Therapy regimen 10 | 1
  Other treatment: Therapy regimen 13: number analyzed (Participants) | 23
  Other treatment: Therapy regimen 13 | 1
  Other treatment: Therapy regimen 18: number analyzed (Participants) | 23
  Other treatment: Therapy regimen 18 | 5
  Other treatment: Therapy regimen 22: number analyzed (Participants) | 23
  Other treatment: Therapy regimen 22 | 2
  Other treatment: Therapy regimen 16: number analyzed (Participants) | 23
  Other treatment: Therapy regimen 16 | 1
  Other treatment: Therapy regimen 4: number analyzed (Participants) | 23
  Other treatment: Therapy regimen 4 | 1

20. Secondary Outcome: Group 2, RRHL: Percentage of Non-ASCT Participants for Whom Treatment is Palliative
Time Frame: as for outcome 10
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 55
percentage of participants
  Palliative at Frontline: number analyzed (Participants) | 39
  Palliative at Frontline | 2.6
  Palliative at Relapse | 43.6

21. Secondary Outcome: Group 2, RRHL: Percentage of Non-ASCT Participants Receiving Positron Emission Tomography (PET) or Computed Tomography (CT) at Each Line of Treatment Pathway
Time Frame: as for outcome 10
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 118
percentage of participants
  PET or PET-CT scan at Baseline | 31.4
  PET or PET-CT scan at Frontline | 59.3
  PET or PET-CT scan at Relapse | 50

22. Secondary Outcome: Group 2, RRHL: Percentage of Non-ASCT Participants Receiving RT at Each Line of Treatment Pathway
Time Frame: as for outcome 10
Population: as for outcome 4
Measure: Number; unit: percentage of participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 201
percentage of participants
  RT at Frontline | 17.4
  RT at Relapse | 22.9

23. Secondary Outcome: Group 2, RRHL: Median Frequency of PET or PET-CT Scan Assessment for Non-ASCT Participants
Time Frame: as for outcome 10
Population: as for outcome 15
Measure: Median (Full Range); unit: scans
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 70
scans
  Frequency of PET or PET-CT Scan at Baseline: number analyzed (Participants) | 37
  Frequency of PET or PET-CT Scan at Baseline | 1.0 [1.0 to 2.0]
  Frequency of PET or PET-CT Scan at Frontline | 1.0 [1.0 to 3.0]
  Frequency of PET or PET-CT Scan at Relapse: number analyzed (Participants) | 59
  Frequency of PET or PET-CT Scan at Relapse | 1.0 [1.0 to 9.0]

24. Secondary Outcome: Group 2, RRHL: Median Number of Treatment Cycles Received in Each Treatment Regimen at Each Line of Treatment in Non-ASCT Participants
Description: Therapy regimens were numbered as 1: ABVD; 3: Stanford V; 6: C-MOPP; 7: DHAP; 11: IGEV; 19: Bendamustine; 4: BEACOPP; 13: MINE; 14: CHOP; 24: Other; 8: ESHAP; 9: Gemcitabine + Carboplatin + Dexamethasone (GCD); 10: ICE; 17: Rituximab; 18: Brentuximab vedotin; 15: CVP; 2: ABVD followed by Escalated BEACOPP; 22: Nivolumab; 16: GVD; 21: Lenalidomide; 24: Other.
Time Frame: From initiation of first treatment until first documentation of relapse/PD/until date of death( or date when participant was last alive), whichever occurred first (observed retrospectively from 2010 until date of data collection [up to 9 years 10 months])
Population: as for outcome 15
Measure: Median (Full Range); unit: cycles
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 161
cycles
  Frontline: Therapy regimen 1 | 6.0 [1.0 to 8.0]
  Frontline: Therapy regimen 3: number analyzed (Participants) | 1
  Frontline: Therapy regimen 3 | 6.0 [6.0 to 6.0]
  Frontline: Therapy regimen 6: number analyzed (Participants) | 1
  Frontline: Therapy regimen 6 | 6.0 [6.0 to 6.0]
  Frontline: Therapy regimen 7: number analyzed (Participants) | 4
  Frontline: Therapy regimen 7 | 3.0 [1.0 to 4.0]
  Frontline: Therapy regimen 11: number analyzed (Participants) | 1
  Frontline: Therapy regimen 11 | 4.0 [4.0 to 4.0]
  Frontline: Therapy regimen 18: number analyzed (Participants) | 1
  Frontline: Therapy regimen 18 | 3.0 [3.0 to 3.0]
  Frontline: Therapy regimen 4: number analyzed (Participants) | 16
  Frontline: Therapy regimen 4 | 6.5 [1.0 to 8.0]
  Frontline: Therapy regimen 14: number analyzed (Participants) | 3
  Frontline: Therapy regimen 14 | 6.0 [6.0 to 6.0]
  Frontline: Therapy regimen 15: number analyzed (Participants) | 1
  Frontline: Therapy regimen 15 | 7.0 [7.0 to 7.0]
  Frontline: Therapy regimen 2: number analyzed (Participants) | 6
  Frontline: Therapy regimen 2 | 7.0 [6.0 to 8.0]
  Frontline: Therapy regimen 24: number analyzed (Participants) | 16
  Frontline: Therapy regimen 24 | 3.0 [1.0 to 7.0]
  Second line: Therapy regimen 1: number analyzed (Participants) | 13
  Second line: Therapy regimen 1 | 4.0 [1.0 to 6.0]
  Second line: Therapy regimen 6: number analyzed (Participants) | 3
  Second line: Therapy regimen 6 | 5.0 [4.0 to 6.0]
  Second line: Therapy regimen 7: number analyzed (Participants) | 23
  Second line: Therapy regimen 7 | 2.0 [1.0 to 4.0]
  Second line: Therapy regimen 8: number analyzed (Participants) | 21
  Second line: Therapy regimen 8 | 2.0 [1.0 to 6.0]
  Second line: Therapy regimen 9: number analyzed (Participants) | 1
  Second line: Therapy regimen 9 | 2.0 [2.0 to 2.0]
  Second line: Therapy regimen 10: number analyzed (Participants) | 18
  Second line: Therapy regimen 10 | 3.0 [1.0 to 8.0]
  Second line: Therapy regimen 11: number analyzed (Participants) | 7
  Second line: Therapy regimen 11 | 4.0 [1.0 to 4.0]
  Second line: Therapy regimen 13: number analyzed (Participants) | 7
  Second line: Therapy regimen 13 | 4.0 [1.0 to 6.0]
  Second line: Therapy regimen 24: number analyzed (Participants) | 39
  Second line: Therapy regimen 24 | 3.0 [1.0 to 12.0]
  Second line: Therapy regimen 17: number analyzed (Participants) | 2
  Second line: Therapy regimen 17 | 3.0 [2.0 to 4.0]
  Second line: Therapy regimen 18: number analyzed (Participants) | 1
  Second line: Therapy regimen 18 | 6.0 [6.0 to 6.0]
  Second line: Therapy regimen 19: number analyzed (Participants) | 1
  Second line: Therapy regimen 19 | 2.0 [2.0 to 2.0]
  Second line: Therapy regimen 4: number analyzed (Participants) | 13
  Second line: Therapy regimen 4 | 4.0 [1.0 to 7.0]
  Second line: Therapy regimen 14: number analyzed (Participants) | 5
  Second line: Therapy regimen 14 | 3.0 [1.0 to 6.0]
  Second line: Therapy regimen 15: number analyzed (Participants) | 1
  Second line: Therapy regimen 15 | 5.0 [5.0 to 5.0]
  Second line: Therapy regimen 2: number analyzed (Participants) | 5
  Second line: Therapy regimen 2 | 6.0 [6.0 to 6.0]
  Third line: Therapy regimen 1: number analyzed (Participants) | 3
  Third line: Therapy regimen 1 | 3.0 [1.0 to 6.0]
  Third line: Therapy regimen 7: number analyzed (Participants) | 4
  Third line: Therapy regimen 7 | 4.0 [2.0 to 6.0]
  Third line: Therapy regimen 8: number analyzed (Participants) | 3
  Third line: Therapy regimen 8 | 2.0 [2.0 to 3.0]
  Third line: Therapy regimen 9: number analyzed (Participants) | 2
  Third line: Therapy regimen 9 | 4.5 [3.0 to 6.0]
  Third line: Therapy regimen 10: number analyzed (Participants) | 8
  Third line: Therapy regimen 10 | 3.5 [2.0 to 8.0]
  Third line: Therapy regimen 11: number analyzed (Participants) | 11
  Third line: Therapy regimen 11 | 2.0 [1.0 to 3.0]
  Third line: Therapy regimen 13: number analyzed (Participants) | 3
  Third line: Therapy regimen 13 | 6.0 [1.0 to 6.0]
  Third line: Therapy regimen 18: number analyzed (Participants) | 3
  Third line: Therapy regimen 18 | 2.0 [2.0 to 4.0]
  Third line: Therapy regimen 17: number analyzed (Participants) | 1
  Third line: Therapy regimen 17 | 12.0 [12.0 to 12.0]
  Third line: Therapy regimen 22: number analyzed (Participants) | 1
  Third line: Therapy regimen 22 | 43.0 [43.0 to 43.0]
  Third line: Therapy regimen 4: number analyzed (Participants) | 2
  Third line: Therapy regimen 4 | 3.5 [2.0 to 5.0]
  Third line: Therapy regimen 24: number analyzed (Participants) | 23
  Third line: Therapy regimen 24 | 3.0 [1.0 to 6.0]
  Other treatments: Therapy regimen 6: number analyzed (Participants) | 1
  Other treatments: Therapy regimen 6 | 1.0 [1.0 to 1.0]
  Other treatments: Therapy regimen 8: number analyzed (Participants) | 1
  Other treatments: Therapy regimen 8 | 2.0 [2.0 to 2.0]
  Other treatments: Therapy regimen 10: number analyzed (Participants) | 1
  Other treatments: Therapy regimen 10 | 4.0 [4.0 to 4.0]
  Other treatments: Therapy regimen 13: number analyzed (Participants) | 1
  Other treatments: Therapy regimen 13 | 6.0 [6.0 to 6.0]
  Other treatments: Therapy regimen 18: number analyzed (Participants) | 5
  Other treatments: Therapy regimen 18 | 6.0 [4.0 to 7.0]
  Other treatments: Therapy regimen 22: number analyzed (Participants) | 2
  Other treatments: Therapy regimen 22 | 12.0 [1.0 to 23.0]
  Other treatments: Therapy regimen 16: number analyzed (Participants) | 1.0
  Other treatments: Therapy regimen 16 | 4.0 [4.0 to 4.0]
  Other treatments: Therapy regimen 4: number analyzed (Participants) | 1
  Other treatments: Therapy regimen 4 | 5.0 [5.0 to 5.0]
  Other treatments: Therapy regimen 24: number analyzed (Participants) | 17
  Other treatments: Therapy regimen 24 | 6.0 [1.0 to 17.0]

25. Secondary Outcome: Group 2, RRHL: Duration of Each Line of Treatment in Non-ASCT Participants
Time Frame: as for outcome 24
Population: as for outcome 15
Measure: Median (Full Range); unit: months
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 201
months
  Frontline Treatment | 5.4 [0.5 to 12.4]
  Second line Treatment: number analyzed (Participants) | 157
  Second line Treatment | 2.2 [0.0 to 8.5]
  Third line Treatment: number analyzed (Participants) | 64
  Third line Treatment | 2.1 [0.0 to 31.6]
  Other Treatment: number analyzed (Participants) | 19
  Other Treatment | 9.7 [0.1 to 44.8]

26. Secondary Outcome: Group 2, RRHL: Percentage of Non-ASCT Participants Categorized Based on Dose Delays in Each Treatment Regimen at Each Line of Treatment
Description: Therapy regimens were numbered as 1: ABVD; 3: Stanford V; 6: C-MOPP; 7: DHAP; 11: IGEV; 4: BEACOPP; 14: CHOP; 15: CVP; 2: ABVD followed by Escalated BEACOPP; 24: Other; 8: ESHAP; 9: GCD; 10: ICE; 13: MINE; 17: Rituximab; 18: Brentuximab vedotin; 19: Bendamustine; 22: Nivolumab. More than one line of treatment or therapy was selected for each participant
Time Frame: as for outcome 10
Population: as for outcome 15
Measure: Number; unit: percentage of participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 161
percentage of participants
  Frontline: Therapy regimen 1 | 14.3
  Frontline: Therapy regimen 3: number analyzed (Participants) | 1
  Frontline: Therapy regimen 3 | 0.0
  Frontline: Therapy regimen 6: number analyzed (Participants) | 1
  Frontline: Therapy regimen 6 | 0.0
  Frontline: Therapy regimen 7: number analyzed (Participants) | 4
  Frontline: Therapy regimen 7 | 0.0
  Frontline: Therapy regimen 11: number analyzed (Participants) | 1
  Frontline: Therapy regimen 11 | 0.0
  Frontline: Therapy regimen 18: number analyzed (Participants) | 1
  Frontline: Therapy regimen 18 | 0.0
  Frontline: Therapy regimen 4: number analyzed (Participants) | 16
  Frontline: Therapy regimen 4 | 6.3
  Frontline: Therapy regimen 15: number analyzed (Participants) | 1
  Frontline: Therapy regimen 15 | 0.0
  Frontline: Therapy regimen 14: number analyzed (Participants) | 3
  Frontline: Therapy regimen 14 | 0.0
  Frontline: Therapy regimen 2: number analyzed (Participants) | 5
  Frontline: Therapy regimen 2 | 0.0
  Frontline: Therapy regimen 24: number analyzed (Participants) | 16
  Frontline: Therapy regimen 24 | 12.5
  Second line: Therapy regimen 1: number analyzed (Participants) | 13
  Second line: Therapy regimen 1 | 2.06
  Second line: Therapy regimen 6: number analyzed (Participants) | 3
  Second line: Therapy regimen 6 | 0.0
  Second line: Therapy regimen 7: number analyzed (Participants) | 23
  Second line: Therapy regimen 7 | 4.3
  Second line: Therapy regimen 8: number analyzed (Participants) | 21
  Second line: Therapy regimen 8 | 0.0
  Second line: Therapy regimen 9: number analyzed (Participants) | 1
  Second line: Therapy regimen 9 | 0.0
  Second line: Therapy regimen 10: number analyzed (Participants) | 18
  Second line: Therapy regimen 10 | 5.6
  Second line: Therapy regimen 11: number analyzed (Participants) | 7
  Second line: Therapy regimen 11 | 14.3
  Second line: Therapy regimen 13: number analyzed (Participants) | 7
  Second line: Therapy regimen 13 | 42.9
  Second line: Therapy regimen 17: number analyzed (Participants) | 2
  Second line: Therapy regimen 17 | 0.0
  Second line: Therapy regimen 18: number analyzed (Participants) | 1
  Second line: Therapy regimen 18 | 0.0
  Second line: Therapy regimen 19: number analyzed (Participants) | 1
  Second line: Therapy regimen 19 | 0.0
  Second line: Therapy regimen 14: number analyzed (Participants) | 5
  Second line: Therapy regimen 14 | 0.0
  Second line: Therapy regimen 15: number analyzed (Participants) | 1
  Second line: Therapy regimen 15 | 0.0
  Second line: Therapy regimen 2: number analyzed (Participants) | 5
  Second line: Therapy regimen 2 | 0.0
  Second line: Therapy regimen 24: number analyzed (Participants) | 38
  Second line: Therapy regimen 24 | 5.3
  Third line: Therapy regimen 1: number analyzed (Participants) | 3
  Third line: Therapy regimen 1 | 33.3
  Third line: Therapy regimen 7: number analyzed (Participants) | 4
  Third line: Therapy regimen 7 | 0.0
  Third line: Therapy regimen 8: number analyzed (Participants) | 3
  Third line: Therapy regimen 8 | 0.0
  Third line: Therapy regimen 9: number analyzed (Participants) | 2
  Third line: Therapy regimen 9 | 50.0
  Third line: Therapy regimen 10: number analyzed (Participants) | 8
  Third line: Therapy regimen 10 | 0.0
  Third line: Therapy regimen 11: number analyzed (Participants) | 11
  Third line: Therapy regimen 11 | 0.0
  Third line: Therapy regimen 13: number analyzed (Participants) | 3
  Third line: Therapy regimen 13 | 33.3
  Third line: Therapy regimen 17: number analyzed (Participants) | 1
  Third line: Therapy regimen 17 | 0.0
  Third line: Therapy regimen 18: number analyzed (Participants) | 3
  Third line: Therapy regimen 18 | 0.0
  Third line: Therapy regimen 22: number analyzed (Participants) | 1
  Third line: Therapy regimen 22 | 0.0
  Third line: Therapy regimen 4: number analyzed (Participants) | 2
  Third line: Therapy regimen 4 | 0.0
  Third line: Therapy regimen 24: number analyzed (Participants) | 24
  Third line: Therapy regimen 24 | 12.5
  Other treatment: Therapy regimen 6: number analyzed (Participants) | 1
  Other treatment: Therapy regimen 6 | 0.0
  Other treatment: Therapy regimen 8: number analyzed (Participants) | 1
  Other treatment: Therapy regimen 8 | 0.0
  Other treatment: Therapy regimen 10: number analyzed (Participants) | 1
  Other treatment: Therapy regimen 10 | 0.0
  Other treatment: Therapy regimen 13: number analyzed (Participants) | 1
  Other treatment: Therapy regimen 13 | 0.0
  Other treatment: Therapy regimen 18: number analyzed (Participants) | 5
  Other treatment: Therapy regimen 18 | 0.0
  Other treatment: Therapy regimen 22: number analyzed (Participants) | 2
  Other treatment: Therapy regimen 22 | 0.0
  Other treatment: Therapy regimen 16: number analyzed (Participants) | 1
  Other treatment: Therapy regimen 16 | 0.0
  Other treatment: Therapy regimen 4: number analyzed (Participants) | 1
  Other treatment: Therapy regimen 4 | 100.0
  Other treatment: Therapy regimen 24: number analyzed (Participants) | 18
  Other treatment: Therapy regimen 24 | 11.1

27. Secondary Outcome: Group 2, RRHL: Time From Relapse (After Frontline Treatment) to First Treatment Post-relapse in Non-ASCT Participants
Time Frame: From relapse after frontline treatment to first treatment post-relapse or until the date of death (or the date when the participant was last known to be alive) (observed retrospectively from 2010 until date of data collection [up to 9 years 10 months])
Population: as for outcome 4
Measure: Median (Full Range); unit: days
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 61
days | 24.0 [1.0 to 902.0]

28. Secondary Outcome: Group 2, RRHL: Time to Initiation of Each Subsequent Treatment, From Relapse and Completion of Previous Treatment in Non-ASCT Participants
Time Frame: From both relapse and from completion of previous treatment to initiation of each subsequent treatment (observed retrospectively from 2010 until date of data collection [up to 9 years 10 months])
Population: as for outcome 15
Measure: Median (Full Range); unit: days
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 17
days
  From end of 1st treatment post 1st relapse to subsequent treatment | 33.0 [1.0 to 148.0]
  From end of 2nd treatment post 1st relapse to subsequent treatment: number analyzed (Participants) | 8
  From end of 2nd treatment post 1st relapse to subsequent treatment | 36.5 [1.0 to 561.0]

29. Secondary Outcome: Group 2, RRHL: Number of Participants With Non-ASCT Assessed for RT Type, Site Received at Frontline
Time Frame: as for outcome 10
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 39
Participants
  RT Type: Whole body | 1
  RT Type: Involved-field | 19
  RT Type: Involved-site | 9
  RT Type: Involved-node | 10
  RT Site: Abdominal nodes | 2
  RT Site: Axillary nodes | 3
  RT Site: Breast | 2
  RT Site: Inguinal nodes | 3
  RT Site: Liver | 1
  RT Site: Mediastinal nodes | 13
  RT Site: Neck nodes | 7
  RT Site: Para-iliac nodes | 1
  RT Site: Pelvic nodes | 1
  RT Site: Soft tissue | 1
  RT Site: Other | 5

30. Secondary Outcome: Group 2, RRHL: Number of Participants With Non-ASCT Assessed for RT Type, Site at Relapse/ Refractory
Time Frame: as for outcome 10
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 55
Participants
  RT Type: Whole body | 0
  RT Type: Involved-field | 24
  RT Type: Involved-site | 20
  RT Type: Involved-node | 10
  RT Type: Other | 1
  RT Site: Abdominal nodes | 2
  RT Site: Axillary nodes | 4
  RT Site: Bone lesions | 8
  RT Site: Brain | 1
  RT Site: Cervix | 1
  RT Site: Inguinal nodes | 2
  RT Site: Mediastinal nodes | 17
  RT Site: Neck nodes | 9
  RT Site: Para-iliac nodes | 1
  RT Site: Pelvic nodes | 3
  RT Site: Supraclavicular nodes | 2
  RT Site: Other | 5

31. Secondary Outcome: Group 2, RRHL: Total Dose of Radiotherapies in Non-ASCT Participants
Time Frame: as for outcome 10
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: Gray
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 31
Gray
  Frontline: number analyzed (Participants) | 23
  Frontline | 36.0 (9.77)
  Relapse/refractory | 30.5 (10.37)

32. Secondary Outcome: Group 2, RRHL: Number of PET or CT Scan Assessments
Time Frame: as for outcome 10
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: scans
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 70
scans
  Baseline: number analyzed (Participants) | 37
  Baseline | 1.1 (0.23)
  Frontline | 1.4 (0.57)
  Relapse: number analyzed (Participants) | 59
  Relapse | 2.0 (1.58)

33. Secondary Outcome: Group 2, RRHL: Number of Participants Categorized Based on Various Chemotherapeutic Regimen and Therapies Used in Participants Undergoing ASCT
Description: Therapy regimens were numbered as 8: ESHAP; 10: ICE; 11: IGEV; 12: Mini-BEAM; 18: Brentuximab vedotin; 19: Bendamustine; 16: GVD; 24: Other. Conditioning regimens are BEAM (Carmustine + Etoposide + Cytarabine + Melphalan), CBV (cyclophosphamide + Carmustine + vp16) BeEAM (bendamustine) and Gemcitabine/Busulfan/Melphalan.
Time Frame: as for outcome 10
Population: The FAS included all participants who were eligible for RRHL group including the common participants in both the groups, and who were undergoing ASCT. Here number analyzed "n" are the participants who were evaluable for the outcome measure at given categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 222
Participants
  Salvage Regimens: Pre-SCT, Therapy regimen 8 | 1
  Salvage Regimens: Pre-SCT, Therapy regimen 10 | 2
  Salvage Regimens: Pre-SCT, Therapy regimen 11 | 1
  Salvage Regimens: Pre-SCT, Therapy regimen 12 | 5
  Salvage Regimens: Pre-SCT, Therapy regimen 18 | 3
  Salvage Regimens: Pre-SCT, Therapy regimen 19 | 1
  Salvage Regimens: Pre-SCT, Therapy regimen 16 | 1
  Salvage Regimens: Pre-SCT, Therapy regimen 24 | 23
  Salvage Regimens: Post-SCT, Therapy regimen 10 | 1
  Salvage Regimens: Post-SCT, Therapy regimen 11 | 1
  Salvage Regimens: Post-SCT, Therapy regimen 18 | 3
  Salvage Regimens: Post-SCT, Therapy regimen 19 | 1
  Salvage Regimens: Post-SCT, Therapy regimen 24 | 2
  Conditioning Regimens: BEAM: number analyzed (Participants) | 216
  Conditioning Regimens: BEAM | 132
  Conditioning Regimens: CBV: number analyzed (Participants) | 216
  Conditioning Regimens: CBV | 22
  Conditioning Regimens: BeEAM: number analyzed (Participants) | 216
  Conditioning Regimens: BeEAM | 6
  Conditioning Regimens: Gemcitabine/Bu/Mel: number analyzed (Participants) | 216
  Conditioning Regimens: Gemcitabine/Bu/Mel | 1
  Conditioning Regimens: Other: number analyzed (Participants) | 216
  Conditioning Regimens: Other | 55
  Conditioning Regimens: Unknown: number analyzed (Participants) | 216
  Conditioning Regimens: Unknown | 3
  Consolidation Therapy : Post -SCT | 4

34. Secondary Outcome: Group 2, RRHL: Number of Participants Categorized Based on With Known Risk Factors for Relapse Post ASCT in Participants Undergoing ASCT
Description: Known risk factors for relapse after ASCT included time to first relapse less than or equal to (<=) 3 months, stage IV disease at relapse, bulky disease >=5 centimeter (cm) at relapse, extranodal disease, inadequate response to salvage chemotherapy (partial remission [PR] or PET positivity), performance status (eastern Cooperative oncology group [ECOG]) >=1. The ECOG assessment used a 3-point scale, including scores of 0 (fully active/able to carry on all pre-disease activities without restriction), 1 (restricted in physically strenuous activity but ambulatory/able to carry out light or sedentary work), or 2 (ambulatory for more than 50% of waking hours and capable of all self care but unable to carry out any work activities).
Time Frame: as for outcome 10
Population: as for outcome 33
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 222
Participants
  Time to first relapse <=3 months: number analyzed (Participants) | 147
  Time to first relapse <=3 months | 19
  Stage IV disease at relapse | 81
  Bulky disease >=5 cm at relapse: number analyzed (Participants) | 218
  Bulky disease >=5 cm at relapse | 47
  Extranodal disease | 83
  Inadequate response to salvage chemotherapy: number analyzed (Participants) | 196
  Inadequate response to salvage chemotherapy | 63
  Performance status (ECOG) >=1: number analyzed (Participants) | 143
  Performance status (ECOG) >=1 | 73

35. Secondary Outcome: Group 2, RRHL: Median Number of Cycles Associated With Each Salvage Regimen in Participants Undergoing ASCT
Description: Therapy regimens were numbered as 1: ABVD; 6: C-MOPP; 7: DHAP; 8: ESHAP; 9: GCD; 10: ICE; 11: IGEV; 12: Mini-BEAM; 13: Eto + Ifosfamide + Mesna + Mitoxantrone (MINE); 18: Brentuximab vedotin; 19: Bendamustine; 22: Nivolumab; 16: GVD; 4: BEACOPP; 14: CHOP; 2: ABVD + Escalated BEACOPP; 24: Other.
Time Frame: as for outcome 10
Population: The FAS included all participants who were eligible for RRHL group including the common participants in both the groups, and who were undergoing ASCT. Here "overall number of participants" analyzed are those who were evaluable for this outcome measure. Here number analyzed "n" are the participants who were evaluable for the outcome measure at given categories.
Measure: Median (Full Range); unit: cycles
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 80
cycles
  Therapy regimen 1: number analyzed (Participants) | 9
  Therapy regimen 1 | 3.0 [1.0 to 8.0]
  Therapy regimen 6: number analyzed (Participants) | 2
  Therapy regimen 6 | 5.5 [3.0 to 8.0]
  Therapy regimen 7: number analyzed (Participants) | 43
  Therapy regimen 7 | 3.0 [1.0 to 6.0]
  Therapy regimen 8 | 3.0 [1.0 to 4.0]
  Therapy regimen 9: number analyzed (Participants) | 3
  Therapy regimen 9 | 2.0 [1.0 to 4.0]
  Therapy regimen 10: number analyzed (Participants) | 45
  Therapy regimen 10 | 3.0 [1.0 to 6.0]
  Therapy regimen 11: number analyzed (Participants) | 40
  Therapy regimen 11 | 3.0 [1.0 to 4.0]
  Therapy regimen 12: number analyzed (Participants) | 10
  Therapy regimen 12 | 1.0 [1.0 to 5.0]
  Therapy regimen 13: number analyzed (Participants) | 9
  Therapy regimen 13 | 5.0 [1.0 to 6.0]
  Therapy regimen 17: number analyzed (Participants) | 1
  Therapy regimen 17 | 8.0 [8.0 to 8.0]
  Therapy regimen 18: number analyzed (Participants) | 29
  Therapy regimen 18 | 6.0 [2.5 to 16.0]
  Therapy regimen 19: number analyzed (Participants) | 15
  Therapy regimen 19 | 4.0 [1.0 to 9.0]
  Therapy regimen 22: number analyzed (Participants) | 4
  Therapy regimen 22 | 6.5 [5.0 to 8.0]
  Therapy regimen 23: number analyzed (Participants) | 1
  Therapy regimen 23 | 21.0 [21.0 to 21.0]
  Therapy regimen 16: number analyzed (Participants) | 8
  Therapy regimen 16 | 3.0 [2.0 to 6.0]
  Therapy regimen 4: number analyzed (Participants) | 7
  Therapy regimen 4 | 4.0 [2.0 to 4.0]
  Therapy regimen 14: number analyzed (Participants) | 2
  Therapy regimen 14 | 1.0 [1.0 to 1.0]
  Therapy regimen 2: number analyzed (Participants) | 1
  Therapy regimen 2 | 2.0 [2.0 to 2.0]
  Therapy regimen 24: number analyzed (Participants) | 68
  Therapy regimen 24 | 2.3 [1.0 to 16.0]

36. Secondary Outcome: Group 2, RRHL: Percentage of Participants Receiving Consolidation Therapy Post-ASCT in Participants Undergoing ASCT
Time Frame: as for outcome 10
Population: The FAS included all participants who were eligible for RRHL group including the common participants in both the groups, and who were undergoing ASCT.
Measure: Number; unit: percentage of participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 222
percentage of participants | 1.4

37. Secondary Outcome: Group 2, RRHL: Median Duration of Treatment for Consolidation Therapies Used in Participants Undergoing ASCT
Time Frame: as for outcome 10
Population: The FAS included all participants who were eligible for RRHL group including the common participants in both the groups, and who were undergoing ASCT. Here "overall number of participants" analyzed are those who received consolidation therapy post-SCT.
Measure: Median (Full Range); unit: months
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 4
months | 11.1 [6.3 to 14.5]

38. Secondary Outcome: Group 2, RRHL: Number of Participants Categorized Based on Source of ASCT Procedures in Participants Undergoing ASCT
Time Frame: as for outcome 10
Population: The FAS included all participants who were eligible for RRHL group including the common participants in both the groups, and who were undergoing ASCT. Here "overall number of participants" analyzed are those who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 219
Participants
  Bone marrow | 36
  Peripheral | 182

39. Secondary Outcome: Group 2, RRHL: Median Time From Relapse (After End of Frontline Treatment) to ASCT in Participants Undergoing ASCT
Time Frame: as for outcome 10
Population: as for outcome 38
Measure: Median (Full Range); unit: days
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 82
days | 182.5 [12.0 to 1021.0]

40. Secondary Outcome: Group 2, RRHL: CD34+ Count Administered in Participants Undergoing ASCT
Time Frame: as for outcome 10
Population: as for outcome 38
Measure: Mean (Standard Deviation); unit: cells per kilogram
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 93
cells per kilogram | 211.2 (248.65)

41. Secondary Outcome: Group 2, RRHL: Time From ASCT to First Relapse in Participants Who Relapse After ASCT
Time Frame: as for outcome 10
Population: The FAS included all participants who were eligible for RRHL group including common participants, and who relapsed after ASCT.
Measure: Median (Full Range); unit: months
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 63
months | 9.9 [2.1 to 78.4]

42. Secondary Outcome: Group 2, RRHL: Number of Participants Categorized Based on Post-ASCT Regimens Received at Each Line of Treatment in Participants Who Relapse After ASCT
Description: Therapy regimens were numbered as 1: ABVD; 7: DHAP; 10: ICE; 11: IGEV; 4: BEACOPP; 2: ABVD followed by Escalated BEACOPP; 8: ESHAP; 12: Mini-BEAM; 13: MINE; 18: Brentuximab vedotin; 22: Nivolumab; 23: Pembrolizumab; 16: GVD, 9: GCD; 24: other; 19: Bendamustine; 14: CHOP; 17: Rituximab.
Time Frame: as for outcome 10
Population: The FAS included all participants who were eligible for RRHL group including common participants, and who relapsed after ASCT. Here number analyzed "n" are the participants who were evaluable for the outcome measure at given categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 63
Participants
  Frontline: Therapy regimen 1 | 57
  Frontline: Therapy regimen 7 | 1
  Frontline: Therapy regimen 10 | 1
  Frontline: Therapy regimen 11 | 1
  Frontline: Therapy regimen 4 | 4
  Frontline: Therapy regimen 2 | 2
  Frontline: Therapy regimen 24 | 3
  Second line: Therapy regimen 7: number analyzed (Participants) | 61
  Second line: Therapy regimen 7 | 9
  Second line: Therapy regimen 8: number analyzed (Participants) | 61
  Second line: Therapy regimen 8 | 28
  Second line: Therapy regimen 10: number analyzed (Participants) | 61
  Second line: Therapy regimen 10 | 10
  Second line: Therapy regimen 11: number analyzed (Participants) | 61
  Second line: Therapy regimen 11 | 4
  Second line: Therapy regimen 12: number analyzed (Participants) | 61
  Second line: Therapy regimen 12 | 1
  Second line: Therapy regimen 13: number analyzed (Participants) | 61
  Second line: Therapy regimen 13 | 2
  Second line: Therapy regimen 18: number analyzed (Participants) | 61
  Second line: Therapy regimen 18 | 1
  Second line: Therapy regimen 4: number analyzed (Participants) | 61
  Second line: Therapy regimen 4 | 4
  Second line: Therapy regimen 24: number analyzed (Participants) | 61
  Second line: Therapy regimen 24 | 5
  Third line: Therapy regimen 7: number analyzed (Participants) | 55
  Third line: Therapy regimen 7 | 2
  Third line: Therapy regimen 8: number analyzed (Participants) | 55
  Third line: Therapy regimen 8 | 3
  Third line: Therapy regimen 9: number analyzed (Participants) | 55
  Third line: Therapy regimen 9 | 3
  Third line: Therapy regimen 10: number analyzed (Participants) | 55
  Third line: Therapy regimen 10 | 6
  Third line: Therapy regimen 11: number analyzed (Participants) | 55
  Third line: Therapy regimen 11 | 9
  Third line: Therapy regimen 12: number analyzed (Participants) | 55
  Third line: Therapy regimen 12 | 3
  Third line: Therapy regimen 13: number analyzed (Participants) | 55
  Third line: Therapy regimen 13 | 1
  Third line: Therapy regimen 18: number analyzed (Participants) | 55
  Third line: Therapy regimen 18 | 9
  Third line: Therapy regimen 22: number analyzed (Participants) | 55
  Third line: Therapy regimen 22 | 1
  Third line: Therapy regimen 23: number analyzed (Participants) | 55
  Third line: Therapy regimen 23 | 1
  Third line: Therapy regimen 16: number analyzed (Participants) | 55
  Third line: Therapy regimen 16 | 4
  Third line: Therapy regimen 4: number analyzed (Participants) | 55
  Third line: Therapy regimen 4 | 1
  Third line: Therapy regimen 24: number analyzed (Participants) | 55
  Third line: Therapy regimen 24 | 13
  Pre-SCT: Therapy regimen 10: number analyzed (Participants) | 16
  Pre-SCT: Therapy regimen 10 | 2
  Pre-SCT: Therapy regimen 12: number analyzed (Participants) | 16
  Pre-SCT: Therapy regimen 12 | 3
  Pre-SCT: Therapy regimen 18: number analyzed (Participants) | 16
  Pre-SCT: Therapy regimen 18 | 2
  Pre-SCT: Therapy regimen 19: number analyzed (Participants) | 16
  Pre-SCT: Therapy regimen 19 | 1
  Pre-SCT: Therapy regimen 14: number analyzed (Participants) | 16
  Pre-SCT: Therapy regimen 14 | 1
  Pre-SCT: Therapy regimen 24: number analyzed (Participants) | 16
  Pre-SCT: Therapy regimen 24 | 9
  Post-SCT: Therapy regimen 18: number analyzed (Participants) | 2
  Post-SCT: Therapy regimen 18 | 2
  Other treatment: Therapy regimen 7: number analyzed (Participants) | 27
  Other treatment: Therapy regimen 7 | 1
  Other treatment: Therapy regimen 9: number analyzed (Participants) | 27
  Other treatment: Therapy regimen 9 | 1
  Other treatment: Therapy regimen 10: number analyzed (Participants) | 27
  Other treatment: Therapy regimen 10 | 2
  Other treatment: Therapy regimen 11: number analyzed (Participants) | 27
  Other treatment: Therapy regimen 11 | 1
  Other treatment: Therapy regimen 17: number analyzed (Participants) | 27
  Other treatment: Therapy regimen 17 | 1
  Other treatment: Therapy regimen 18: number analyzed (Participants) | 27
  Other treatment: Therapy regimen 18 | 7
  Other treatment: Therapy regimen 19: number analyzed (Participants) | 27
  Other treatment: Therapy regimen 19 | 7
  Other treatment: Therapy regimen 22: number analyzed (Participants) | 27
  Other treatment: Therapy regimen 22 | 5
  Other treatment: Therapy regimen 23: number analyzed (Participants) | 27
  Other treatment: Therapy regimen 23 | 2
  Other treatment: Therapy regimen 16: number analyzed (Participants) | 27
  Other treatment: Therapy regimen 16 | 1
  Other treatment: Therapy regimen 4: number analyzed (Participants) | 27
  Other treatment: Therapy regimen 4 | 1
  Other treatment: Therapy regimen 24: number analyzed (Participants) | 27
  Other treatment: Therapy regimen 24 | 15

43. Secondary Outcome: Group 2, RRHL: Percentage of Participants Who Relapse After ASCT Categorized Based on Palliative Therapy Regimens
Description: Therapy regimens were numbered as 9: GVD; 10: ICE; 11: IGEV; 12: Mini-BEAM; 18: Brentuximab vedotin; 19: Bendamustine; 22: Nivolumab.
Time Frame: as for outcome 10
Population: The FAS included all participants who were eligible for RRHL group including common participants, and who relapsed after ASCT. Here "overall number of participants" analyzed are those who were evaluable for this outcome measure.
Measure: Number; unit: percentage of participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 8
percentage of participants
  Therapy regimen 9 | 12.5
  Therapy regimen 10 | 12.5
  Therapy regimen 11 | 12.5
  Therapy regimen 12 | 12.5
  Therapy regimen 18 | 12.5
  Therapy regimen 19 | 12.5
  Therapy regimen 22 | 12.5
  Other | 75.0

44. Secondary Outcome: Group 2, RRHL: Number of Cycles Received at Each Line of Treatment for Each Treatment Regimen in Participants Who Relapse After ASCT
Description: Therapy regimens were numbered as 1: ABVD; 7: DHAP; 10: ICE; 11: IGEV; 4: BEACOPP; 2: ABVD followed by Escalated BEACOPP; 8: ESHAP; 12: Mini-BEAM; 13: MINE; 18: Brentuximab vedotin; 9: GCD; 22: Nivolumab; 23: Pembrolizumab; 16: GVD.
Time Frame: as for outcome 10
Population: as for outcome 42
Measure: Median (Full Range); unit: cycles
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 63
cycles
  Frontline: Therapy regimen 1: number analyzed (Participants) | 57
  Frontline: Therapy regimen 1 | 6.0 [2.0 to 8.0]
  Frontline: Therapy regimen 7: number analyzed (Participants) | 1
  Frontline: Therapy regimen 7 | 2.0 [2.0 to 2.0]
  Frontline: Therapy regimen 10: number analyzed (Participants) | 1
  Frontline: Therapy regimen 10 | 2.0 [2.0 to 2.0]
  Frontline: Therapy regimen 11: number analyzed (Participants) | 1
  Frontline: Therapy regimen 11 | 2.0 [2.0 to 2.0]
  Frontline: Therapy regimen 4: number analyzed (Participants) | 4
  Frontline: Therapy regimen 4 | 6.0 [6.0 to 8.0]
  Frontline: Therapy regimen 2: number analyzed (Participants) | 2
  Frontline: Therapy regimen 2 | 7.0 [6.0 to 8.0]
  Frontline: Therapy regimen 24: number analyzed (Participants) | 3
  Frontline: Therapy regimen 24 | 2.0 [1.0 to 4.0]
  Second line: Therapy regimen 7: number analyzed (Participants) | 9
  Second line: Therapy regimen 7 | 2.0 [1.0 to 6.0]
  Second line: Therapy regimen 8: number analyzed (Participants) | 28
  Second line: Therapy regimen 8 | 3.0 [1.0 to 6.0]
  Second line: Therapy regimen 10: number analyzed (Participants) | 10
  Second line: Therapy regimen 10 | 3.0 [1.0 to 3.0]
  Second line: Therapy regimen 11: number analyzed (Participants) | 4
  Second line: Therapy regimen 11 | 3.0 [3.0 to 4.0]
  Second line: Therapy regimen 12: number analyzed (Participants) | 1
  Second line: Therapy regimen 12 | 1.0 [1.0 to 1.0]
  Second line: Therapy regimen 13: number analyzed (Participants) | 2
  Second line: Therapy regimen 13 | 3.5 [1.0 to 6.0]
  Second line: Therapy regimen 18: number analyzed (Participants) | 1
  Second line: Therapy regimen 18 | 3.0 [3.0 to 3.0]
  Second line: Therapy regimen 4: number analyzed (Participants) | 4
  Second line: Therapy regimen 4 | 4.0 [2.0 to 6.0]
  Second line: Therapy regimen 24: number analyzed (Participants) | 5
  Second line: Therapy regimen 24 | 4.0 [2.0 to 8.0]
  Third line: Therapy regimen 7: number analyzed (Participants) | 2
  Third line: Therapy regimen 7 | 1.5 [1.0 to 2.0]
  Third line: Therapy regimen 8: number analyzed (Participants) | 3
  Third line: Therapy regimen 8 | 2.0 [2.0 to 3.0]
  Third line: Therapy regimen 9: number analyzed (Participants) | 3
  Third line: Therapy regimen 9 | 6.0 [2.0 to 6.0]
  Third line: Therapy regimen 10: number analyzed (Participants) | 6
  Third line: Therapy regimen 10 | 3.0 [1.0 to 6.0]
  Third line: Therapy regimen 11: number analyzed (Participants) | 9
  Third line: Therapy regimen 11 | 3.0 [1.0 to 4.0]
  Third line: Therapy regimen 12: number analyzed (Participants) | 3
  Third line: Therapy regimen 12 | 2.0 [1.0 to 4.0]
  Third line: Therapy regimen 13: number analyzed (Participants) | 1
  Third line: Therapy regimen 13 | 6.0 [6.0 to 6.0]
  Third line: Therapy regimen 18: number analyzed (Participants) | 9
  Third line: Therapy regimen 18 | 5.0 [3.0 to 16.0]
  Third line: Therapy regimen 22: number analyzed (Participants) | 1
  Third line: Therapy regimen 22 | 8.0 [8.0 to 8.0]
  Third line: Therapy regimen 23: number analyzed (Participants) | 1
  Third line: Therapy regimen 23 | 1.0 [1.0 to 1.0]
  Third line: Therapy regimen 16: number analyzed (Participants) | 4
  Third line: Therapy regimen 16 | 3.0 [3.0 to 6.0]
  Third line: Therapy regimen 4: number analyzed (Participants) | 1
  Third line: Therapy regimen 4 | 3.0 [3.0 to 3.0]
  Pre-SCT: Therapy regimen 10: number analyzed (Participants) | 2
  Pre-SCT: Therapy regimen 10 | 2.0 [2.0 to 2.0]
  Pre-SCT: Therapy regimen 12: number analyzed (Participants) | 3
  Pre-SCT: Therapy regimen 12 | 1.0 [1.0 to 1.0]
  Pre-SCT: Therapy regimen 18: number analyzed (Participants) | 2
  Pre-SCT: Therapy regimen 18 | 7.5 [5.0 to 10.0]
  Pre-SCT: Therapy regimen 19 | 6.0 [6.0 to 6.0]
  Pre-SCT: Therapy regimen 14 | 1.0 [1.0 to 1.0]
  Pre-SCT: Therapy regimen 24: number analyzed (Participants) | 9
  Pre-SCT: Therapy regimen 24 | 1.0 [1.0 to 1.0]
  Post-SCT: Therapy regimen 18: number analyzed (Participants) | 2
  Post-SCT: Therapy regimen 18 | 9.0 [6.0 to 12.0]
  Other treatment: Therapy regimen 7 | 3.0 [3.0 to 3.0]
  Other treatment: Therapy regimen 9 | 4.0 [4.0 to 4.0]
  Other treatment: Therapy regimen 10: number analyzed (Participants) | 2
  Other treatment: Therapy regimen 10 | 2.5 [2.0 to 3.0]
  Other treatment: Therapy regimen 11 | 4.0 [4.0 to 4.0]
  Other treatment: Therapy regimen 17 | 8.0 [8.0 to 8.0]
  Other treatment: Therapy regimen 18: number analyzed (Participants) | 7
  Other treatment: Therapy regimen 18 | 12.0 [2.0 to 16.0]
  Other treatment: Therapy regimen 19: number analyzed (Participants) | 7
  Other treatment: Therapy regimen 19 | 4.0 [2.0 to 9.0]
  Other treatment: Therapy regimen 22: number analyzed (Participants) | 5
  Other treatment: Therapy regimen 22 | 7.0 [5.0 to 26.0]
  Other treatment: Therapy regimen 23: number analyzed (Participants) | 2
  Other treatment: Therapy regimen 23 | 23.0 [21.0 to 25.0]
  Other treatment: Therapy regimen 16 | 2.0 [2.0 to 2.0]
  Other treatment: Therapy regimen 4 | 2.0 [2.0 to 2.0]
  Other treatment: Therapy regimen 24: number analyzed (Participants) | 15
  Other treatment: Therapy regimen 24 | 4.0 [1.0 to 16.0]

45. Secondary Outcome: Group 2, RRHL: Duration of Each Line of Treatment for Participants Who Relapse After ASCT
Time Frame: as for outcome 10
Population: as for outcome 42
Measure: Median (Full Range); unit: months
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 63
months
  Frontline Treatment | 5.9 [0.0 to 11.9]
  Second line Treatment: number analyzed (Participants) | 61
  Second line Treatment | 2.0 [0.0 to 9.4]
  Third line Treatment: number analyzed (Participants) | 53
  Third line Treatment | 2.0 [0.1 to 13.2]
  Pre-SCT Treatment: number analyzed (Participants) | 16
  Pre-SCT Treatment | 0.2 [0.0 to 6.0]
  Post-SCT Treatment: number analyzed (Participants) | 2
  Post-SCT Treatment | 7.2 [5.6 to 8.8]
  Other Treatment: number analyzed (Participants) | 27
  Other Treatment | 4.0 [0.7 to 18.5]

46. Secondary Outcome: Group 2, RRHL: Time From ASCT to First Treatment After Relapse in Participants Who Relapse After ASCT
Time Frame: as for outcome 10
Population: as for outcome 43
Measure: Median (Full Range); unit: months
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 52
months | 16.0 [2.9 to 53.8]

47. Secondary Outcome: Group 2, RRHL: Time to Initiation of Each Subsequent Treatment, From ASCT and From Completion of Previous Treatment in Participants Who Relapse From ASCT
Time Frame: as for outcome 10
Population: The FAS included all participants who were eligible for RRHL group including common participants, and who relapsed after ASCT. Here "overall number of participants" analyzed are those who were evaluable for this outcome measure. Here number analyzed "n" are the participants who were evaluable for the outcome measure at given categories.
Measure: Median (Full Range); unit: months
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 52
months
  From ASCT to 1st treatment | 16.0 [2.9 to 53.8]
  From ASCT to 2nd treatment: number analyzed (Participants) | 20
  From ASCT to 2nd treatment | 19.1 [9.1 to 87.4]
  From ASCT to 3rd treatment: number analyzed (Participants) | 7
  From ASCT to 3rd treatment | 28.1 [17.7 to 90.9]
  From completion of 1st treatment to next treatment: number analyzed (Participants) | 20
  From completion of 1st treatment to next treatment | 63.0 [25.0 to 1596.0]
  From completion of 2nd treatment to next treatment: number analyzed (Participants) | 7
  From completion of 2nd treatment to next treatment | 87.0 [59.0 to 544.0]

48. Secondary Outcome: Group 2, RRHL: Percentage of Participants Who Received PET-CT Scan, CT Scan and Radiotherapy at Each Stage of the Treatment Pathway in Participants Who Relapse After ASCT
Description: Data for PET-CT scan and CT scans were assessed for baseline, frontline and relapse/or refractory, and radiotherapy was assessed for frontline and relapse/refractory, as planned.
Time Frame: as for outcome 10
Population: as for outcome 42
Measure: Number; unit: percentage of participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 63
percentage of participants
  PET-CT scan: Baseline: number analyzed (Participants) | 55
  PET-CT scan: Baseline | 23.6
  PET-CT scan: Frontline: number analyzed (Participants) | 55
  PET-CT scan: Frontline | 54.5
  PET-CT scan: Relapse and /or refractory: number analyzed (Participants) | 55
  PET-CT scan: Relapse and /or refractory | 60.0
  CT scan: Baseline: number analyzed (Participants) | 48
  CT scan: Baseline | 47.9
  CT scan: Frontline: number analyzed (Participants) | 48
  CT scan: Frontline | 60.4
  CT scan: Relapse and /or refractory: number analyzed (Participants) | 48
  CT scan: Relapse and /or refractory | 70.8
  Radiotherapy: Frontline | 22.2
  Radiotherapy: Relapse/refractory | 36.5

49. Secondary Outcome: Group 2, RRHL: Mean Frequency of PET or PET-CT Scan Assessments for Participants Who Relapse After ASCT
Description: Data for PET-CT scan and CT scans were assessed for baseline, frontline and relapse or refractory, as planned.
Time Frame: as for outcome 10
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: scans
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 34
scans
  PET or PET-CT scan: Baseline: number analyzed (Participants) | 13
  PET or PET-CT scan: Baseline | 1.0 (0.00)
  PET or PET-CT scan: Frontline: number analyzed (Participants) | 30
  PET or PET-CT scan: Frontline | 2.0 (1.26)
  PET or PET-CT scan: Relapse /refractory: number analyzed (Participants) | 33
  PET or PET-CT scan: Relapse /refractory | 5.6 (3.62)
  CT Scan: Baseline: number analyzed (Participants) | 23
  CT Scan: Baseline | 1.0 (0.21)
  CT Scan: Frontline: number analyzed (Participants) | 29
  CT Scan: Frontline | 2.6 (2.26)
  CT Scan: Relapse/refractory | 4.3 (4.37)

50. Secondary Outcome: Group 2, RRHL: Number of Participants With Types of Radiotherapies Received at Frontline and at Relapse/Refractory in Participants Who Relapse After ASCT
Time Frame: From initial diagnosis and until death or date of data collected, whichever occurred first (observed retrospectively from 2010 until date of data collection [up to 9 years 10 months])
Population: as for outcome 47
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 23
Participants
  Frontline: Whole body: number analyzed (Participants) | 14
  Frontline: Whole body | 1
  Frontline: Involved-field radiotherapy: number analyzed (Participants) | 14
  Frontline: Involved-field radiotherapy | 8
  Frontline: Involved-site radiotherapy: number analyzed (Participants) | 14
  Frontline: Involved-site radiotherapy | 4
  Frontline: Involved-node radiotherapy: number analyzed (Participants) | 14
  Frontline: Involved-node radiotherapy | 2
  Relapse/refractory: Whole body | 1
  Relapse/refractory: Involved-field radiotherapy | 21
  Relapse/refractory: Involved-site radiotherapy | 4
  Relapse/refractory: Involved-node radiotherapy | 3
  Relapse/refractory: Other | 1

51. Secondary Outcome: Group 2, RRHL: Number of Participants Categorized Based on Anatomical Site of Radiotherapies in Participants Who Relapse After ASCT at Frontline and at Relapse/Refractory
Time Frame: as for outcome 10
Population: as for outcome 47
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 23
Participants
  Frontline: Axillary nodes: number analyzed (Participants) | 14
  Frontline: Axillary nodes | 1
  Frontline: Bone lesions: number analyzed (Participants) | 14
  Frontline: Bone lesions | 1
  Frontline: Mediastinal nodes: number analyzed (Participants) | 14
  Frontline: Mediastinal nodes | 4
  Frontline: Neck nodes: number analyzed (Participants) | 14
  Frontline: Neck nodes | 2
  Frontline: Other: number analyzed (Participants) | 14
  Frontline: Other | 7
  Relapse/refractory: Abdominal nodes | 4
  Relapse/refractory: Axillary nodes | 4
  Relapse/refractory: Bone lesions | 3
  Relapse/refractory: Mediastinal nodes | 12
  Relapse/refractory: Neck nodes | 5
  Relapse/refractory: Other | 2

52. Secondary Outcome: Group 2, RRHL: Number of Participants Categorized Based on Intent of Treatment of Radiotherapies in Participants Who Relapse After ASCT
Time Frame: as for outcome 10
Population: as for outcome 41
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 63
Participants
  Frontline: Radical/Cure Intent | 14
  Frontline: Other | 1
  Relapse/refractory: Radical/Cure Intent | 23
  Relapse/refractory: Palliative Intent | 5
  Relapse/refractory: Other | 2

53. Secondary Outcome: Group 2, RRHL: Total Dose of Radiotherapies Received at Frontline and Relapse/Refractory in Participants Who Relapse After ASCT
Time Frame: as for outcome 10
Population: as for outcome 47
Measure: Mean (Standard Deviation); unit: Gray
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 20
Gray
  Total Dose of RT at Frontline: number analyzed (Participants) | 12
  Total Dose of RT at Frontline | 32.0 (7.28)
  Total Dose of RT at Relapse/refractory | 33.0 (6.96)

54. Secondary Outcome: Group 2, RRHL: Percentage of Participants Undergoing Subsequent ASCTs and Allogeneic Stem Cell Transplantation (Allo-SCT)
Time Frame: as for outcome 10
Population: as for outcome 43
Measure: Number; unit: percentage of participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 20
percentage of participants
  Undergoing subsequent ASCTs | 38.1
  Undergoing allo-SCT | 4.8

55. Secondary Outcome: Group 2, RRHL: Group 2, RRHL: Median Number of ASCTs for Each Participant Who Relapse After ASCT
Time Frame: as for outcome 10
Population: as for outcome 41
Measure: Median (Full Range); unit: ASCTs
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 63
ASCTs | 1.0 [1.0 to 2.0]

56. Secondary Outcome: Group 1, cHL: Median PFS
Description: PFS was defined as time from initiation of frontline regimen to first documentation of relapse or disease progression or death, censored at date of most recent follow-up/contact. PD was defined as any new lesion or increase by >= 50% of previously involved site from nadir, and was evaluated based on IWG criteria (Cheson et al 2007). Median PFS was estimated using the Kaplan-Meier method.
Time Frame: From initiation of frontline regimen to first documentation of relapse/PD/until date of death (or date when participant was last alive), whichever occurred first (observed retrospectively from 2010 until date of data collection [up to 9 years 10 months])
Population: The FAS included all participants who were eligible for cHL group including the common participants in both the groups.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 1: cHL
Number analyzed (Participants) | 1598
months | NA [NA to NA] — Median, lower and upper limit of 95% confidence interval (CI) could not be calculated because insufficient number of participants had events.

57. Secondary Outcome: Group 1, cHL: Number of Participants Based on Best Clinical Response Post Completion of Frontline Treatment
Description: Best clinical response as complete remission (CR), partial remission (PR), stable disease (SD), or PD was evaluated based on IWG criteria (Cheson et al 2007). CR was the disappearance of all evidence of disease. PR was the regression of measurable disease and no new sites. SD was defined by failure to achieve CR, PR, or PD. PD was defined as any new lesion or increase by >=50% of previously involved sites from nadir.
Time Frame: From post completion of frontline treatment until the date of death (or the date when the participant was last known to be alive) (observed retrospectively from 2010 until date of data collection [up to 9 years 10 months])
Population: The FAS included all participants who were eligible for cHL group including the common participants in both the groups.
Measure: Number; unit: participants
Arm/Group | Group 1: cHL
Number analyzed (Participants) | 1598
participants
  CR | 968
  PR | 356
  SD | 80
  PD | 109
  Other | 85

58. Secondary Outcome: Group 2, RRHL: Number of Participants With Best Clinical Response Post Completion of Each Line of Treatment
Description: Best clinical response as CR, PR, SD, or PD was evaluated based on IWG criteria (Cheson et al 2007). CR was the disappearance of all evidence of disease. PR was the regression of measurable disease and no new sites. SD was defined by failure to achieve CR, PR, or PD. PD was defined as any new lesion or increase by >=50% of previously involved sites from nadir.
Time Frame: as for outcome 57
Population: The FAS included all participants who were eligible for RRHL group including the common participants in both the groups. Here number analyzed "n" are the participants who were evaluable for the outcome measure at given categories.
Measure: Number; unit: participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 426
participants
  Frontline: CR | 131
  Frontline: PR | 133
  Frontline: SD | 40
  Frontline: PD | 98
  Frontline: Other | 24
  Second line: CR: number analyzed (Participants) | 374
  Second line: CR | 107
  Second line: PR: number analyzed (Participants) | 374
  Second line: PR | 113
  Second line: SD: number analyzed (Participants) | 374
  Second line: SD | 32
  Second line: PD: number analyzed (Participants) | 374
  Second line: PD | 80
  Second line: Other: number analyzed (Participants) | 374
  Second line: Other | 42
  Third line: CR: number analyzed (Participants) | 178
  Third line: CR | 46
  Third line: PR: number analyzed (Participants) | 178
  Third line: PR | 38
  Third line: SD: number analyzed (Participants) | 178
  Third line: SD | 22
  Third line: PD: number analyzed (Participants) | 178
  Third line: PD | 48
  Third line: Other | 24
  Pre-SCT: CR: number analyzed (Participants) | 50
  Pre-SCT: CR | 14
  Pre-SCT: PR: number analyzed (Participants) | 50
  Pre-SCT: PR | 12
  Pre-SCT: SD: number analyzed (Participants) | 50
  Pre-SCT: SD | 2
  Pre-SCT: PD: number analyzed (Participants) | 50
  Pre-SCT: PD | 4
  Post-SCT: CR: number analyzed (Participants) | 10
  Post-SCT: CR | 5
  Pre-SCT: Other: number analyzed (Participants) | 50
  Pre-SCT: Other | 18
  Post-SCT: PR: number analyzed (Participants) | 10
  Post-SCT: PR | 1
  Post-SCT: SD: number analyzed (Participants) | 10
  Post-SCT: SD | 1
  Post-SCT: PD: number analyzed (Participants) | 10
  Post-SCT: PD | 2
  Post-SCT: Other: number analyzed (Participants) | 10
  Post-SCT: Other | 1
  Other line: CR: number analyzed (Participants) | 69
  Other line: CR | 17
  Other line: PR: number analyzed (Participants) | 69
  Other line: PR | 17
  Other line: SD: number analyzed (Participants) | 69
  Other line: SD | 10
  Other line: PD: number analyzed (Participants) | 69
  Other line: PD | 15
  Other line: Other | 10

59. Secondary Outcome: Mean Duration of Best Response
Description: Duration of best response was defined as the time from when the criteria for response (CR or PR) were met to first documentation of relapse or disease progression, and was evaluated based on IWG criteria (Cheson et al 2007). CR was the disappearance of all evidence of disease. PR was the regression of measurable disease and no new sites. PD was defined as any new lesion or increase by >=50% of previously involved sites from nadir.
Time Frame: From CR or PR until first documentation of relapse or disease progression or until the date of death (or the date when the participant was last known to be alive) (observed retrospectively from 2010 until date of data collection [up to 9 years 10 months])
Population: The FAS included all participants who were eligible for cHL or RRHL group including the common participants in both the groups. Here "overall number of participants" analyzed are those who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 1: cHL | Group 2: RRHL
Number analyzed (Participants) | 1452 | 298
months | NA [NA to NA] — Median, lower and upper limit of 95% CI could not be calculated because insufficient number of participants had an event. | 51.08 [27.07 to NA] — The upper 95% CI was not achieved due to high censoring rate.

60. Secondary Outcome: Median Overall Survival (OS)
Description: Median OS was defined as the time from diagnosis of cHL to death(Group 1)/ time from first relapse after frontline therapy to death (Group 2), censored at date of most recent follow-up/contact.
Time Frame: From initial diagnosis until the date of death (or date when the participant was alive) (Group 1); From first relapse after frontline therapy to death (Group 2) (observed retrospectively from 2010 until date of data collection [up to 9 years 10 months])
Population: as for outcome 59
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 1: cHL | Group 2: RRHL
Number analyzed (Participants) | 1598 | 249
months | NA [NA to NA] — Median, lower and upper limit of 95% CI could not be calculated because insufficient number of participants had an event. | NA [NA to NA] — Median, lower and upper limit of 95% CI could not be calculated because insufficient number of participants had an event.

61. Secondary Outcome: Group 1, cHL: Overall Survival Rate After Diagnosis at 1 and 5 Years
Description: Percentage of participants who were alive at 1 and 5 years after diagnosis in cHL participants are reported. 5 year overall survival data were reported only for participants who had >5 year observation periods.
Time Frame: At 1 year and 5 years after diagnosis (observed retrospectively from 2010 until date of data collection [up to 9 years 10 months])
Population: The FAS included all participants who were eligible for cHL group including the common participants in both the groups.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 1: cHL
Number analyzed (Participants) | 1598
percentage of participants
  At 1 year | 95.65 [94.52 to 96.56]
  At 5 years | 84.74 [82.75 to 86.52]

62. Secondary Outcome: Group 2, RRHL: Overall Survival Rate at 1 and 5 Years
Description: Percentage of participants who were alive at 1 and 5 years after diagnosis in RRHL participants are reported. 5 year overall survival data were reported only for participants who had >5 year observation periods.
Time Frame: At 1 year and 5 years after relapse (observed retrospectively from 2010 until date of data collection [up to 9 years 10 months])
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 249
percentage of participants
  At 1 year | 89.15 [84.48 to 92.48]
  At 5 years | 70.68 [64.10 to 76.28]

63. Secondary Outcome: Group 1, cHL: Number of Participants Who Had Inpatient Hospital Admissions, Emergency Room Visits, and Outpatient Visits by Healthcare Professionals Related to HL
Time Frame: as for outcome 10
Population: The FAS included all participants who were eligible for cHL group including common participants in both the groups.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: cHL
Number analyzed (Participants) | 1598
Participants
  Inpatient Hospital Admissions | 864
  Emergency Room Visits | 357
  Outpatient Visits | 1135

64. Secondary Outcome: Group 1, cHL: Number of Participants Categorized Based on Reasons for Inpatient Hospital Admissions Related to HL
Time Frame: as for outcome 10
Population: The FAS included all participants who were eligible for cHL group including common participants in both the groups, and who had HL inpatient hospitalizations.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: cHL
Number analyzed (Participants) | 864
Participants
  Chemotherapy | 563
  Radiotherapy | 39
  Stem cell transplant | 146
  Adverse event | 287
  Unknown | 37
  Other | 384

65. Secondary Outcome: Group 1, cHL: Mean Overall Length of Stay and Length of Stay by Unit/Ward for Inpatient Hospital Admissions Related to HL
Description: Length of stay by unit or ward included general, high dependency/intermediate, intensive care unit, bone marrow transplant unit, and emergency visits.
Time Frame: as for outcome 10
Population: The FAS included all participants who were eligible for cHL group including common participants in both the groups, and who had HL inpatient hospitalizations. Here number analyzed "n" are the participants who were evaluable for the outcome measure at given categories.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group 1: cHL
Number analyzed (Participants) | 864
days
  Overall length of stay | 15.1 (41.02)
  Length of stay by unit/ward: General: number analyzed (Participants) | 789
  Length of stay by unit/ward: General | 13.2 (41.86)
  Length of stay by unit/ward: High dependency/intermediate: number analyzed (Participants) | 56
  Length of stay by unit/ward: High dependency/intermediate | 20.2 (17.29)
  Length of stay by unit/ward: Intensive Care Unit: number analyzed (Participants) | 48
  Length of stay by unit/ward: Intensive Care Unit | 28.0 (26.14)
  Length of stay by unit/ward: Bone marrow transplant unit: number analyzed (Participants) | 100
  Length of stay by unit/ward: Bone marrow transplant unit | 32.7 (39.70)

66. Secondary Outcome: Group 1, cHL: Number of Participants Categorized Based on Episodes of RT Received, Type of Scan or Procedure, and Who Received Granulocyte-colony Stimulating Factor (G-CSF) or High-cost Medicines and Pegylated G-CSF Related to HL
Time Frame: as for outcome 10
Population: The FAS included all participants who were eligible for cHL group including common participants in both the groups. Here number analyzed "n" are the participants who were evaluable for the outcome measure at given categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1: cHL
Number analyzed (Participants) | 1598
Participants
  RT received | 357
  Scan/procedure: Chest x-Ray: number analyzed (Participants) | 1597
  Scan/procedure: Chest x-Ray | 427
  Scan/procedure: Magnetic resonance imaging (MRI): number analyzed (Participants) | 1597
  Scan/procedure: Magnetic resonance imaging (MRI) | 92
  Scan/procedure: Needle biopsy: number analyzed (Participants) | 1597
  Scan/procedure: Needle biopsy | 273
  Scan/procedure: Bone scan: number analyzed (Participants) | 1597
  Scan/procedure: Bone scan | 19
  Scan/procedure: Bone marrow aspiration: number analyzed (Participants) | 1597
  Scan/procedure: Bone marrow aspiration | 997
  Scan/procedure: Flow cytometry: number analyzed (Participants) | 1597
  Scan/procedure: Flow cytometry | 61
  Scan/procedure: Other scan procedures: number analyzed (Participants) | 1597
  Scan/procedure: Other scan procedures | 315
  Received G-CSF/ other high cost medications | 794
  Received Pegylated G-CSF | 143

67. Secondary Outcome: Group 1, cHL: Mean Number of Courses of Treatment With G-CSF/Pegylated G-CSF or Other High-cost Medicines Related to HL Treatment
Time Frame: as for outcome 10
Population: The FAS included all participants who were eligible for cHL group including common participants in both the groups. Here "overall number of participants" analyzed are those who were evaluable for this outcome measure. Here number analyzed "n" are the participants who were evaluable for the outcome measure at given categories.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group 1: cHL
Number analyzed (Participants) | 792
days
  Courses: G-CSF treatment/other high cost medicines | 5.6 (6.99)
  Courses: Pegylated G-CSF: number analyzed (Participants) | 143
  Courses: Pegylated G-CSF | 2.5 (2.99)

68. Secondary Outcome: Group 2, RRHL: Number of Participants Who Had Inpatient Hospital Admissions, Emergency Room Visits, and Outpatient Visits by Healthcare Professional Related to HL for Salvage Therapy and ASCT
Description: Each participant had more than one category presented for salvage therapy and ASCT.
Time Frame: as for outcome 10
Population: The FAS included all participants who were eligible for RRHL group including common participants in both the groups. Here "overall number of participants" analyzed are those who were evaluable for this outcome measure. Here number analyzed "n" are the participants who were evaluable for the outcome measure at given categories.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 333
Participants
  Salvage Therapy: Inpatient Hospital Admissions | 175
  Salvage Therapy: Emergency Room Visits | 44
  Salvage Therapy: Outpatient Visits | 185
  ASCT: Inpatient Hospital Admissions: number analyzed (Participants) | 188
  ASCT: Inpatient Hospital Admissions | 5
  ASCT: Emergency Room Visits: number analyzed (Participants) | 188
  ASCT: Emergency Room Visits | 2
  ASCT: Outpatient Visits: number analyzed (Participants) | 188
  ASCT: Outpatient Visits | 4

69. Secondary Outcome: Group 2, RRHL: Number of Participants Categorized Based on Reasons for Inpatient Hospital Admissions Related to HL for Salvage Therapy and ASCT
Description: Each participant had more than one category presented for salvage therapy and ASCT.
Time Frame: as for outcome 10
Population: as for outcome 68
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 175
Participants
  Salvage Therapy: Chemotherapy | 144
  Salvage Therapy: Radiotherapy | 6
  Salvage Therapy: Stem cell transplant | 50
  Salvage Therapy: Adverse event | 36
  Salvage Therapy: Unknown | 6
  Salvage Therapy: Other | 51
  ASCT: Chemotherapy: number analyzed (Participants) | 5
  ASCT: Chemotherapy | 2
  ASCT: Adverse event: number analyzed (Participants) | 5
  ASCT: Adverse event | 3

70. Secondary Outcome: Group 2, RRHL: Mean Overall Length of Stay and Length of Stay by Unit/Ward for Inpatient Hospital Admissions Related to HL for Salvage Therapy and ASCT
Description: Length of stay by unit or ward included general, high dependency/intermediate, intensive care unit, bone marrow transplant unit, and emergency visits. Each participant had more than one category presented for salvage therapy and ASCT.
Time Frame: as for outcome 10
Population: The FAS included all participants who were eligible for RRHL group including common participants in both the groups. Here number analyzed "n" are the participants who were evaluable for the outcome measure at given categories.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 426
days
  Salvage Therapy: Overall length of stay | 13.6 (16.30)
  Salvage Therapy: General: number analyzed (Participants) | 158
  Salvage Therapy: General | 11.4 (15.79)
  Salvage Therapy: High dependency/intermediate: number analyzed (Participants) | 12
  Salvage Therapy: High dependency/intermediate | 25.8 (18.24)
  Salvage Therapy: Intensive Care Unit: number analyzed (Participants) | 2
  Salvage Therapy: Intensive Care Unit | 13.0 (7.07)
  Salvage Therapy: Bone marrow transplant unit: number analyzed (Participants) | 32
  Salvage Therapy: Bone marrow transplant unit | 25.8 (10.08)
  ASCT: Overall length of stay: number analyzed (Participants) | 5
  ASCT: Overall length of stay | 7.8 (4.54)
  ASCT: General: number analyzed (Participants) | 3
  ASCT: General | 4.9 (1.23)
  ASCT: High dependency/intermediate: number analyzed (Participants) | 2
  ASCT: High dependency/intermediate | 10.5 (6.36)
  ASCT: Intensive Care Unit: number analyzed (Participants) | 1
  ASCT: Intensive Care Unit | 18.0 (NA) — Standard deviation could not be calculated because only one participant was evaluable.
  ASCT: Bone marrow transplant unit: number analyzed (Participants) | 0

71. Secondary Outcome: Group 2, RRHL: Number of Participants Categorized Based on Episodes of RT, Type of Scan or Procedure, and Who Received G-CSF or High-cost Medicines Related to HL for Salvage Therapy and ASCT
Description: Each participant had more than one category presented for salvage therapy and ASCT. Scan procedures included chest x-ray, magnetic resonance imaging, needle biopsy, bone scan, bone marrow aspiration, flow cytometry, and other scan procedures.
Time Frame: as for outcome 10
Population: as for outcome 68
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 188
Participants
  Salvage Therapy: Chest x-Ray: number analyzed (Participants) | 117
  Salvage Therapy: Chest x-Ray | 63
  Salvage Therapy: Magnetic resonance imaging: number analyzed (Participants) | 117
  Salvage Therapy: Magnetic resonance imaging | 8
  Salvage Therapy: Needle biopsy: number analyzed (Participants) | 117
  Salvage Therapy: Needle biopsy | 19
  Salvage Therapy: Bone scan: number analyzed (Participants) | 117
  Salvage Therapy: Bone scan | 3
  Salvage Therapy: Bone marrow aspiration: number analyzed (Participants) | 117
  Salvage Therapy: Bone marrow aspiration | 43
  Salvage Therapy: Flow cytometry: number analyzed (Participants) | 117
  Salvage Therapy: Flow cytometry | 4
  Salvage Therapy: Other scan procedures: number analyzed (Participants) | 117
  Salvage Therapy: Other scan procedures | 40
  Salvage Therapy: G-CSF/ other high cost medications: number analyzed (Participants) | 150
  Salvage Therapy: G-CSF/ other high cost medications | 150
  Salvage Therapy: Pegylated G-CSF: number analyzed (Participants) | 146
  Salvage Therapy: Pegylated G-CSF | 17
  ASCT: Chest x-ray: number analyzed (Participants) | 0
  ASCT: Magnetic resonance imaging: number analyzed (Participants) | 0
  ASCT: Needle biopsy: number analyzed (Participants) | 0
  ASCT: Bone scan: number analyzed (Participants) | 0
  ASCT: Bone marrow aspiration: number analyzed (Participants) | 0
  ASCT: Flow cytometry: number analyzed (Participants) | 0
  ASCT: Other scan procedures: number analyzed (Participants) | 0
  ASCT: G-CSF/ other high cost medications | 6
  ASCT: Pegylated G-CSF: number analyzed (Participants) | 6
  ASCT: Pegylated G-CSF | 1

72. Secondary Outcome: Group 2, RRHL: Group 2, RRHL: Mean Number of Courses of Treatment With G-CSF/Pegylated G-CSF or Other High-cost Medicines Related to HL Treatment for Salvage Therapy and ASCT
Time Frame: as for outcome 10
Population: as for outcome 68
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Group 2: RRHL
Number analyzed (Participants) | 150
days
  Salvage Therapy: G-CSF treatment/other high cost medicines | 2.8 (2.78)
  Salvage Therapy: Pegylated G-CSF: number analyzed (Participants) | 17
  Salvage Therapy: Pegylated G-CSF | 2.6 (2.90)
  ASCT: G-CSF treatment/other high cost medicines: number analyzed (Participants) | 6
  ASCT: G-CSF treatment/other high cost medicines | 4.2 (2.64)
  ASCT: Pegylated G-CSF: number analyzed (Participants) | 1
  ASCT: Pegylated G-CSF | 6.0 (NA) — Standard deviation could not be calculated because only one participant was evaluable.

ADVERSE EVENTS:
Time Frame: From initial diagnosis until the date of death (or the date when the participant was last known to be alive) (observed retrospectively from 2010 until date of data collection [up to 9 years 10 months])
Description: At each visit the investigator had to assess any occurrence of adverse events. Participants may report adverse events occurring at any other time during the study. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | Group 1: cHL | Group 2: RRHL
All-Cause Mortality (participants affected / at risk) | 243/1598 | 136/426
Serious Adverse Events (participants affected / at risk) | 303/1598 | 103/426
Other Adverse Events (participants affected / at risk) | 642/1598 | 187/426
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: cHL (N=1598) | Group 2: RRHL (N=426)
Febrile neutropenia (Blood and lymphatic system disorders) | 69 | 25
Neutropenia (Blood and lymphatic system disorders) | 30 | 8
Anaemia (Blood and lymphatic system disorders) | 15 | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 7 | 1
Pancytopenia (Blood and lymphatic system disorders) | 5 | 3
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0
Platelet disorder (Blood and lymphatic system disorders) | 1 | 0
Pneumonia (Infections and infestations) | 33 | 6
Neutropenic sepsis (Infections and infestations) | 8 | 6
Herpes zoster (Infections and infestations) | 7 | 4
Sepsis (Infections and infestations) | 6 | 3
Urinary tract infection (Infections and infestations) | 5 | 2
Septic shock (Infections and infestations) | 4 | 0
Bacteraemia (Infections and infestations) | 3 | 1
Device related infection (Infections and infestations) | 3 | 2
Cellulitis (Infections and infestations) | 2 | 0
Lower respiratory tract infection (Infections and infestations) | 2 | 0
Lung infection (Infections and infestations) | 2 | 2
Upper respiratory tract infection (Infections and infestations) | 2 | 0
Abscess limb (Infections and infestations) | 1 | 0
Acute sinusitis (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 1 | 1
Anal infection (Infections and infestations) | 1 | 0
Appendicitis (Infections and infestations) | 1 | 0
Aspergillus infection (Infections and infestations) | 1 | 0
Bacterial sepsis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Carbuncle (Infections and infestations) | 1 | 0
Catheter site infection (Infections and infestations) | 1 | 1
Clostridial sepsis (Infections and infestations) | 1 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0
Cryptococcosis (Infections and infestations) | 1 | 1
Cystitis (Infections and infestations) | 1 | 0
Device related sepsis (Infections and infestations) | 1 | 1
Endocarditis (Infections and infestations) | 1 | 1
Fungal sepsis (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Herpes simplex (Infections and infestations) | 1 | 0
Herpes virus infection (Infections and infestations) | 1 | 1
Herpes zoster disseminated (Infections and infestations) | 1 | 1
Infection (Infections and infestations) | 1 | 1
Influenza (Infections and infestations) | 1 | 1
Klebsiella sepsis (Infections and infestations) | 1 | 1
Large intestine infection (Infections and infestations) | 1 | 1
Mastoiditis (Infections and infestations) | 1 | 0
Mucormycosis (Infections and infestations) | 1 | 1
Osteomyelitis (Infections and infestations) | 1 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0
Pneumonia chlamydial (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 1
Renal abscess (Infections and infestations) | 1 | 1
Systemic candida (Infections and infestations) | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 1
Klebsiella bacteraemia (Infections and infestations) | 2 | 0
Pyrexia (General disorders) | 46 | 16
Asthenia (General disorders) | 3 | 1
Chest pain (General disorders) | 2 | 0
Mucosal inflammation (General disorders) | 2 | 2
Adverse drug reaction (General disorders) | 1 | 1
Catheter site necrosis (General disorders) | 1 | 0
Death (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 1
Gait disturbance (General disorders) | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 9 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 6 | 0
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Acute lung injury (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Mediastinal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 6 | 1
Nausea (Gastrointestinal disorders) | 3 | 1
Stomatitis (Gastrointestinal disorders) | 3 | 1
Vomiting (Gastrointestinal disorders) | 3 | 1
Abdominal pain (Gastrointestinal disorders) | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 2 | 1
Constipation (Gastrointestinal disorders) | 2 | 2
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Duodenal perforation (Gastrointestinal disorders) | 1 | 0
Duodenitis (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Oesophagitis (Gastrointestinal disorders) | 1 | 1
Rectal prolapse (Gastrointestinal disorders) | 1 | 1
Ascites (Gastrointestinal disorders) | 2 | 0
Neutropenic colitis (Gastrointestinal disorders) | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 5 | 3
Bradycardia (Cardiac disorders) | 2 | 0
Cardiac tamponade (Cardiac disorders) | 2 | 2
Myocardial infarction (Cardiac disorders) | 2 | 0
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Angina pectoris (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 1 | 0
Cardiomyopathy (Cardiac disorders) | 1 | 0
Cardiotoxicity (Cardiac disorders) | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 0
Palpitations (Cardiac disorders) | 1 | 1
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 0
Headache (Nervous system disorders) | 5 | 1
Neuropathy peripheral (Nervous system disorders) | 3 | 1
Dizziness (Nervous system disorders) | 2 | 0
Hemiplegia (Nervous system disorders) | 1 | 0
Monoparesis (Nervous system disorders) | 1 | 0
Myxoedema coma (Nervous system disorders) | 1 | 0
Speech disorder (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 1 | 1
Subdural hygroma (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 0
Tension headache (Nervous system disorders) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 6 | 1
Traumatic lung injury (Injury, poisoning and procedural complications) | 4 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Pneumonitis chemical (Injury, poisoning and procedural complications) | 1 | 0
Radiation mucositis (Injury, poisoning and procedural complications) | 1 | 1
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 2 | 0
Tumour lysis syndrome (Metabolism and nutrition disorders) | 2 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2
Drug hypersensitivity (Immune system disorders) | 3 | 0
Graft versus host disease in gastrointestinal tract (Immune system disorders) | 2 | 2
Acute graft versus host disease (Immune system disorders) | 1 | 1
Graft versus host disease (Immune system disorders) | 1 | 0
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 | 1
Acute graft versus host disease in skin (Immune system disorders) | 1 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myofascial pain syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0
Synovitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Hypotension (Vascular disorders) | 3 | 0
Arterial haemorrhage (Vascular disorders) | 1 | 0
Hypovolaemic shock (Vascular disorders) | 1 | 1
Phlebitis (Vascular disorders) | 1 | 0
Thrombophlebitis superficial (Vascular disorders) | 1 | 0
Blood bilirubin increased (Investigations) | 1 | 0
Ejection fraction decreased (Investigations) | 1 | 1
General physical condition abnormal (Investigations) | 1 | 1
Neutrophil count decreased (Investigations) | 1 | 0
Platelet count decreased (Investigations) | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 2
Cystitis haemorrhagic (Renal and urinary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 2 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0
Diffuse large B-cell lymphoma stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Post transplant lymphoproliferative disorder (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Diplopia (Eye disorders) | 1 | 1
Photophobia (Eye disorders) | 1 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Hypercalcaemia of malignancy (Endocrine disorders) | 1 | 1
Delirium (Psychiatric disorders) | 1 | 1
Vaginal ulceration (Reproductive system and breast disorders) | 1 | 0
Bone marrow failure (Blood and lymphatic system disorders) | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 1
Otitis media (Infections and infestations) | 0 | 1
Multiple organ dysfunction syndrome (General disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Engraftment syndrome (Immune system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1: cHL (N=1598) | Group 2: RRHL (N=426)
Neutropenia (Blood and lymphatic system disorders) | 256 | 80
Leukopenia (Blood and lymphatic system disorders) | 68 | 24
Febrile neutropenia (Blood and lymphatic system disorders) | 56 | 29
Anaemia (Blood and lymphatic system disorders) | 46 | 20
Thrombocytopenia (Blood and lymphatic system disorders) | 27 | 20
Bone marrow failure (Blood and lymphatic system disorders) | 22 | 12
Erythropenia (Blood and lymphatic system disorders) | 5 | 1
Pancytopenia (Blood and lymphatic system disorders) | 3 | 1
Agranulocytosis (Blood and lymphatic system disorders) | 1 | 1
Autoimmune haemolytic anaemia (Blood and lymphatic system disorders) | 1 | 1
Bicytopenia (Blood and lymphatic system disorders) | 1 | 0
Cytopenia (Blood and lymphatic system disorders) | 1 | 1
Eosinophilia (Blood and lymphatic system disorders) | 1 | 0
Haematotoxicity (Blood and lymphatic system disorders) | 1 | 0
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 70 | 24
Vomiting (Gastrointestinal disorders) | 60 | 20
Constipation (Gastrointestinal disorders) | 31 | 8
Stomatitis (Gastrointestinal disorders) | 30 | 13
Diarrhoea (Gastrointestinal disorders) | 28 | 14
Gastrointestinal disorder (Gastrointestinal disorders) | 24 | 11
Abdominal pain (Gastrointestinal disorders) | 14 | 7
Mouth ulceration (Gastrointestinal disorders) | 12 | 2
Abdominal pain upper (Gastrointestinal disorders) | 9 | 3
Dyspepsia (Gastrointestinal disorders) | 6 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 2
Abdominal discomfort (Gastrointestinal disorders) | 4 | 1
Abdominal distension (Gastrointestinal disorders) | 4 | 1
Haemorrhoids (Gastrointestinal disorders) | 4 | 0
Odynophagia (Gastrointestinal disorders) | 4 | 1
Dysphagia (Gastrointestinal disorders) | 3 | 2
Epigastric discomfort (Gastrointestinal disorders) | 2 | 1
Gastritis (Gastrointestinal disorders) | 2 | 0
Proctalgia (Gastrointestinal disorders) | 2 | 1
Proctitis (Gastrointestinal disorders) | 2 | 1
Anal fissure (Gastrointestinal disorders) | 1 | 0
Aphthous ulcer (Gastrointestinal disorders) | 1 | 0
Chronic gastritis (Gastrointestinal disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Dry mouth (Gastrointestinal disorders) | 1 | 1
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 1
Gastritis erosive (Gastrointestinal disorders) | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrointestinal inflammation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 | 0
Gingival bleeding (Gastrointestinal disorders) | 1 | 0
Gingival pain (Gastrointestinal disorders) | 1 | 1
Glossodynia (Gastrointestinal disorders) | 1 | 0
Intestinal cyst (Gastrointestinal disorders) | 1 | 0
Large intestinal stenosis (Gastrointestinal disorders) | 1 | 0
Lip ulceration (Gastrointestinal disorders) | 1 | 2
Oesophagitis (Gastrointestinal disorders) | 1 | 1
Oral mucosal eruption (Gastrointestinal disorders) | 1 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 1
Salivary gland pain (Gastrointestinal disorders) | 1 | 1
Toothache (Gastrointestinal disorders) | 1 | 1
Pneumonia (Infections and infestations) | 18 | 5
Upper respiratory tract infection (Infections and infestations) | 17 | 5
Herpes zoster (Infections and infestations) | 9 | 4
Urinary tract infection (Infections and infestations) | 8 | 3
Influenza (Infections and infestations) | 6 | 1
Sepsis (Infections and infestations) | 6 | 1
Lung infection (Infections and infestations) | 5 | 0
Oral candidiasis (Infections and infestations) | 5 | 1
Pharyngitis (Infections and infestations) | 5 | 1
Sinusitis (Infections and infestations) | 5 | 2
Device related sepsis (Infections and infestations) | 4 | 3
Anal abscess (Infections and infestations) | 3 | 2
Cellulitis (Infections and infestations) | 3 | 1
Folliculitis (Infections and infestations) | 3 | 2
Furuncle (Infections and infestations) | 3 | 0
Nasopharyngitis (Infections and infestations) | 3 | 1
Oesophageal candidiasis (Infections and infestations) | 3 | 0
Clostridium difficile colitis (Infections and infestations) | 2 | 0
Cytomegalovirus infection (Infections and infestations) | 2 | 2
Gastroenteritis (Infections and infestations) | 2 | 4
Genital herpes (Infections and infestations) | 2 | 0
Gingivitis (Infections and infestations) | 2 | 1
Herpes virus infection (Infections and infestations) | 2 | 0
Infection (Infections and infestations) | 2 | 0
Neutropenic sepsis (Infections and infestations) | 2 | 1
Oropharyngeal candidiasis (Infections and infestations) | 2 | 1
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 | 0
Pulmonary tuberculosis (Infections and infestations) | 2 | 0
Respiratory tract infection (Infections and infestations) | 2 | 0
Varicella (Infections and infestations) | 2 | 0
Vascular device infection (Infections and infestations) | 2 | 2
Acute sinusitis (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Bronchitis bacterial (Infections and infestations) | 1 | 0
Bronchopulmonary aspergillosis (Infections and infestations) | 1 | 1
Conjunctivitis (Infections and infestations) | 1 | 0
Conjunctivitis viral (Infections and infestations) | 1 | 1
Device related infection (Infections and infestations) | 1 | 0
Endocarditis (Infections and infestations) | 1 | 1
Epstein-Barr virus infection (Infections and infestations) | 1 | 0
Fungal infection (Infections and infestations) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Genital infection fungal (Infections and infestations) | 1 | 0
Lip infection (Infections and infestations) | 1 | 1
Nail bed infection (Infections and infestations) | 1 | 0
Onychomycosis (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Orchitis (Infections and infestations) | 1 | 0
Otitis media (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 1 | 0
Pathogen resistance (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia cytomegaloviral (Infections and infestations) | 1 | 0
Pneumonia fungal (Infections and infestations) | 1 | 0
Postpartum sepsis (Infections and infestations) | 1 | 1
Rash pustular (Infections and infestations) | 1 | 0
Rhinitis (Infections and infestations) | 1 | 1
Skin candida (Infections and infestations) | 1 | 0
Soft tissue infection (Infections and infestations) | 1 | 0
Staphylococcal bacteraemia (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 1
Tinea infection (Infections and infestations) | 1 | 0
Tinea pedis (Infections and infestations) | 1 | 0
Tonsillitis (Infections and infestations) | 1 | 0
Tracheobronchitis (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Vulvovaginal candidiasis (Infections and infestations) | 1 | 0
Pyrexia (General disorders) | 68 | 45
Fatigue (General disorders) | 31 | 12
Pain (General disorders) | 8 | 4
Malaise (General disorders) | 7 | 2
Oedema peripheral (General disorders) | 7 | 5
Non-cardiac chest pain (General disorders) | 6 | 5
Asthenia (General disorders) | 5 | 1
Chills (General disorders) | 5 | 2
Mucosal inflammation (General disorders) | 5 | 4
Swelling (General disorders) | 3 | 0
Adverse drug reaction (General disorders) | 2 | 0
Chest discomfort (General disorders) | 2 | 0
Peripheral swelling (General disorders) | 2 | 1
Axillary pain (General disorders) | 1 | 1
Catheter site pain (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Extravasation (General disorders) | 1 | 0
Gait disturbance (General disorders) | 1 | 1
Hyperthermia (General disorders) | 1 | 0
Inflammation (General disorders) | 1 | 1
Influenza like illness (General disorders) | 1 | 0
Injection site hypoaesthesia (General disorders) | 1 | 0
Injection site pain (General disorders) | 1 | 0
Sensation of foreign body (General disorders) | 1 | 0
Vessel puncture site pain (General disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 28 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 21 | 7
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 14 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 6
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Organising pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oropharyngeal spasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngeal disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Neuropathy peripheral (Nervous system disorders) | 42 | 7
Headache (Nervous system disorders) | 18 | 6
Dizziness (Nervous system disorders) | 16 | 7
Hypoaesthesia (Nervous system disorders) | 10 | 4
Facial paralysis (Nervous system disorders) | 2 | 0
Neurotoxicity (Nervous system disorders) | 2 | 0
Paraesthesia (Nervous system disorders) | 2 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 0
Cerebellar infarction (Nervous system disorders) | 1 | 1
Lethargy (Nervous system disorders) | 1 | 1
Neuritis (Nervous system disorders) | 1 | 1
Polyneuropathy (Nervous system disorders) | 1 | 1
Somnolence (Nervous system disorders) | 1 | 0
Taste disorder (Nervous system disorders) | 1 | 0
Toxic neuropathy (Nervous system disorders) | 1 | 0
Neutrophil count decreased (Investigations) | 35 | 15
Haemoglobin decreased (Investigations) | 28 | 14
Platelet count decreased (Investigations) | 6 | 5
Weight decreased (Investigations) | 6 | 2
White blood cell count decreased (Investigations) | 4 | 2
Alanine aminotransferase increased (Investigations) | 2 | 0
International normalised ratio increased (Investigations) | 2 | 1
Transaminases increased (Investigations) | 2 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 1
Blood uric acid increased (Investigations) | 1 | 0
Campylobacter test positive (Investigations) | 1 | 0
Cytomegalovirus test (Investigations) | 1 | 1
Ejection fraction decreased (Investigations) | 1 | 0
HIV test positive (Investigations) | 1 | 0
Oxygen saturation decreased (Investigations) | 1 | 0
Serum ferritin increased (Investigations) | 1 | 1
Total lung capacity decreased (Investigations) | 1 | 1
Transaminases abnormal (Investigations) | 1 | 0
Urine analysis normal (Investigations) | 1 | 1
Venous pressure (Investigations) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 13 | 8
Alopecia (Skin and subcutaneous tissue disorders) | 12 | 3
Night sweats (Skin and subcutaneous tissue disorders) | 9 | 3
Rash (Skin and subcutaneous tissue disorders) | 7 | 7
Rash pruritic (Skin and subcutaneous tissue disorders) | 6 | 2
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 6 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 5 | 1
Erythema (Skin and subcutaneous tissue disorders) | 5 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 5 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 4 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 1
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3 | 1
Eczema (Skin and subcutaneous tissue disorders) | 3 | 1
Rash generalised (Skin and subcutaneous tissue disorders) | 3 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 2 | 0
Skin exfoliation (Skin and subcutaneous tissue disorders) | 2 | 1
Skin reaction (Skin and subcutaneous tissue disorders) | 2 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 2 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 1 | 1
Dermatosis (Skin and subcutaneous tissue disorders) | 1 | 0
Generalised erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 | 0
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 1 | 0
Onychomadesis (Skin and subcutaneous tissue disorders) | 1 | 0
Papule (Skin and subcutaneous tissue disorders) | 1 | 1
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 1 | 1
Post inflammatory pigmentation change (Skin and subcutaneous tissue disorders) | 1 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 1 | 0
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 1
Skin discolouration (Skin and subcutaneous tissue disorders) | 1 | 0
Skin toxicity (Skin and subcutaneous tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 12 | 6
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 5
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 7 | 5
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 7 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 2
Pain in jaw (Musculoskeletal and connective tissue disorders) | 2 | 1
Clubbing (Musculoskeletal and connective tissue disorders) | 1 | 0
Enthesopathy (Musculoskeletal and connective tissue disorders) | 1 | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Periostitis (Musculoskeletal and connective tissue disorders) | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 16 | 10
Hypokalaemia (Metabolism and nutrition disorders) | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 2 | 0
Fluid overload (Metabolism and nutrition disorders) | 1 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1
Hypophagia (Metabolism and nutrition disorders) | 1 | 2
Increased appetite (Metabolism and nutrition disorders) | 1 | 0
Iron overload (Metabolism and nutrition disorders) | 1 | 0
Steroid diabetes (Metabolism and nutrition disorders) | 1 | 1
Deep vein thrombosis (Vascular disorders) | 4 | 1
Hot flush (Vascular disorders) | 4 | 1
Orthostatic hypotension (Vascular disorders) | 3 | 1
Thrombophlebitis superficial (Vascular disorders) | 3 | 0
Hypotension (Vascular disorders) | 2 | 0
Jugular vein thrombosis (Vascular disorders) | 2 | 2
Pallor (Vascular disorders) | 2 | 1
Phlebitis (Vascular disorders) | 2 | 1
Thrombophlebitis (Vascular disorders) | 2 | 0
Thrombosis (Vascular disorders) | 2 | 1
Embolism venous (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 1
Varicose vein (Vascular disorders) | 1 | 0
Vasculitis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 9 | 2
Traumatic lung injury (Injury, poisoning and procedural complications) | 3 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0
Gastrointestinal injury (Injury, poisoning and procedural complications) | 1 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 1 | 2
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 1
Joint injury (Injury, poisoning and procedural complications) | 1 | 0
Radiation pneumonitis (Injury, poisoning and procedural complications) | 1 | 0
Transfusion reaction (Injury, poisoning and procedural complications) | 1 | 1
Insomnia (Psychiatric disorders) | 7 | 5
Anxiety (Psychiatric disorders) | 3 | 1
Depression (Psychiatric disorders) | 2 | 0
Bipolar I disorder (Psychiatric disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 1
Delirium (Psychiatric disorders) | 1 | 0
Depressed mood (Psychiatric disorders) | 1 | 0
Drug hypersensitivity (Immune system disorders) | 2 | 2
Graft versus host disease in skin (Immune system disorders) | 2 | 2
Hypersensitivity (Immune system disorders) | 2 | 0
Anaphylactic reaction (Immune system disorders) | 1 | 0
Chronic graft versus host disease (Immune system disorders) | 1 | 1
Chronic graft versus host disease in skin (Immune system disorders) | 1 | 1
Engraftment syndrome (Immune system disorders) | 1 | 0
Graft versus host disease (Immune system disorders) | 1 | 1
Palpitations (Cardiac disorders) | 5 | 3
Angina pectoris (Cardiac disorders) | 2 | 0
Arrhythmia (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Cystitis haemorrhagic (Renal and urinary disorders) | 2 | 0
Dysuria (Renal and urinary disorders) | 2 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 1
Renal impairment (Renal and urinary disorders) | 1 | 0
Renal vascular thrombosis (Renal and urinary disorders) | 1 | 1
Renal vein thrombosis (Renal and urinary disorders) | 1 | 1
Urinary tract disorder (Renal and urinary disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 3 | 3
Hypoacusis (Ear and labyrinth disorders) | 2 | 1
Vertigo (Ear and labyrinth disorders) | 2 | 1
Vision blurred (Eye disorders) | 3 | 2
Macular pigmentation (Eye disorders) | 1 | 0
Swelling of eyelid (Eye disorders) | 1 | 0
Visual acuity reduced (Eye disorders) | 1 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Gastrooesophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Marginal zone lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Ovarian germ cell teratoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gynaecomastia (Reproductive system and breast disorders) | 2 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0
Vulvovaginal pruritus (Reproductive system and breast disorders) | 1 | 0
Hepatic steatosis (Hepatobiliary disorders) | 1 | 1
Hepatitis toxic (Hepatobiliary disorders) | 1 | 0
Hepatotoxicity (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 1 | 1
Hypothyroidism (Endocrine disorders) | 2 | 0
Autoimmune hypothyroidism (Endocrine disorders) | 1 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0
Catheter site rash (General disorders) | 0 | 1
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 0 | 1
Tongue ulceration (Gastrointestinal disorders) | 0 | 1
Bronchiolitis (Infections and infestations) | 0 | 1
Febrile infection (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 0 | 1
Tooth abscess (Infections and infestations) | 0 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Presyncope (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 0 | 1
Dyshidrotic eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Diabetic metabolic decompensation (Metabolism and nutrition disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1
Liver injury (Hepatobiliary disorders) | 0 | 1
Ovarian cyst (Reproductive system and breast disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.

DOCUMENTS (2):
  • Study Protocol (2017-05-04): https://cdn.clinicaltrials.gov/large-docs/71/NCT03327571/Prot_000.pdf
  • Statistical Analysis Plan (2020-02-24): https://cdn.clinicaltrials.gov/large-docs/71/NCT03327571/SAP_001.pdf